Protocol Title: Evaluation of the clinical performance of Daily Disposable Silicone Hydrogel

Multifocal Toric Contact Lenses

Protocol Number: CR-6542

Version: 4.0

Date: 25 March 2024

Investigational products: JJVC Investigational Multifocal Toric Contact Lenses manufactured in Senofilcon A (C3) material with UV blocker and HEV filter

Key Words: Presbyopia, Multifocal, Astigmatism, Daily Wear, Daily Disposable, Dispensing, senofilcon A, logMAR visual acuity, CLUE questionnaire, Single arm

### Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This trial will be conducted in compliance with ISO 14155:2020 Clinical investigation of medical devices for human subjects – Good clinical practice<sup>1</sup>, the Declaration of Helsinki<sup>2</sup>, and all applicable regulatory requirements<sup>3</sup>.

### **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.

| | | CONTENTS<br>FITLE, NUMBER, VERSION AND DATE | 7 |
|---|---|---|---|
| | | AME AND ADDRESS | |
| | | ONITOR | |
| | | D SIGNATURES | |
| | | STORY | |
| | | 71011 | |
| | | USED ABBREVIATIONS, ACRONYMS AND DEFINITION | |
| 1. IN | TRODI | UCTION AND BACKGROUND | 19 |
| 1.1. | Name | e and Descriptions of Investigational Products | 19 |
| 1.2. | Intend | ded Use of Investigational Products | 19 |
| 1.3. | Sumn | nary of Findings from Nonclinical Studies | 19 |
| 1.4. | Sumn | nary of Known Risks and Benefits to Human Subjects | 19 |
| 1.5. | | vant Literature References and Prior Clinical Data Relevant to Pr | |
| • | | | |
| 2. ST | | OBJECTIVES, ENDPOINTS AND HYPOTHESES | |
| 2.1. | Objec | ctives | 21 |
| 2.2. | Endpo | oints | |
| 2.2 | 2.1. | Co-Primary Efficacy Endpoints | |
| 2.2 | 2.2. | Co-Primary Safety Endpoints | |
| | 2.3. | Secondary Efficacy Endpoints | |
| 2.3. | Hypo | theses | |
| 2.3 | 3.1. | Co-Primary Efficacy Hypotheses | 23 |
| 2.3 | 3.2. | Co-Primary Safety Hypotheses | 24 |
| 2.3 | 3.3. | Secondary Efficacy Hypotheses | 24 |
| 3. TA | RGET | ED STUDY POPULATION | |
| 3.1. | Gener | ral Characteristics | 25 |
| 3.2. | Inclus | sion Criteria | 25 |
| 3.3. | Exclu | sion Criteria | 25 |
| 3.4. | Enrol | lment Strategy | 26 |
| 4. ST | UDY I | DESIGN AND RATIONALE | 27 |
| 4.1. | Descr | ription of Study Design | 27 |
| 42 | Study | Design Rationale | 27 |

| 4.3. | Enrollment Target and Study Duration | 27 |
|--------------|-----------------------------------------------------|----|
| 5. TE | ST ARTICLE ALLOCATION AND MASKING | 27 |
| 5.1. | Test Article Allocation | 27 |
| 5.2. | Masking | 28 |
| 5.3. | Procedures for Maintaining and Breaking the Masking | 28 |
| 6. ST | UDY INTERVENTION | 28 |
| 6.1. | Identity of Test Articles. | 28 |
| 6.2. | Ancillary Supplies/Products | 29 |
| 6.3. | Administration of Test Articles | 29 |
| 6.4. | Packaging and Labeling | 30 |
| 6.5. | Storage Conditions | 30 |
| 6.6. | Collection and Storage of Samples | 30 |
| 6.7. | Accountability of Test Articles | 30 |
| 7. ST | UDY EVALUATIONS | 31 |
| 7.1. | Time and Event Schedule | 31 |
| 7.2. | Detailed Study Procedures | 33 |
| VI | SIT 1 | 33 |
| VI | SIT 2 | 41 |
| VI | SIT 3 | 47 |
| FII | NAL EVALUATION | 49 |
| 7.3. | Unscheduled Visits | 50 |
| 7.4. | Laboratory Procedures | 52 |
| 8. SU | BJECTS COMPLETION/WITHDRAWAL | 53 |
| 8.1. | Completion Criteria | 53 |
| 8.2. | Withdrawal/Discontinuation from the Study | 53 |
| 9. PR | E-STUDY AND CONCOMITANT INTERVENTION/MEDICATION | |
| 9.1. | Systemic Medications | 54 |
| | DEVIATIONS FROM THE PROTOCOL | |
| 11. | STUDY TERMINATION | 56 |
| 12. I | PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS | 56 |
| 13. <i>A</i> | ADVERSE EVENTS | 57 |
| 13.1. | Definitions and Classifications. | 57 |
| 13.2. | Assessing Adverse Events | 60 |
| 13 | .2.1. Causality Assessment | 60 |

| 13.2 | 2.2. Severity Assessment | 61 |
|---|---|---|
| 13.3. | Documentation and Follow-Up of Adverse Events | 61 |
| 13.4. | Reporting Adverse Events | 62 |
| 13.4 | 4.1. Reporting Adverse Events to Sponsor | 62 |
| _ | 4.2. Reporting Adverse Events to the Responsible IEC/IRB and Heathorities | |
| 13.5. | Event of Special Interest | 63 |
| 13.6. | Reporting of Pregnancy | 63 |
| 14. S | TATISTICAL METHODS | 64 |
| 14.1. | General Considerations | 64 |
| 14.2. | Sample Size Justification | 64 |
| 14.3. | Analysis Populations | 69 |
| 14.4. | Level of Statistical Significance. | 69 |
| 14.5. | Primary Analysis | 69 |
| 14.5 | 5.1. Co-Primary Efficacy Analyses | 69 |
| 14.5 | 5.2. Co-Primary Safety Analyses | 73 |
| 14.6. | Secondary Analyses | 74 |
| 14.7. | Exploratory Analyses | 77 |
| 14.8. | Interim Analysis | 77 |
| 14.9. | Procedure for Handling Missing Data and Drop-Outs | 77 |
| 14.10. | Procedure for Reporting Deviations from Statistical Plan | 77 |
| 15. D | ATA HANDLING AND RECORD KEEPING/ARCHIVING | 77 |
| 15.1. | Electronic Case Report Form/Data Collection | 77 |
| 15.2. | Subject Record | 78 |
| 15.3. | Trial Registration on ClinicalTrials.gov | 78 |
| 16. D | ATA MANAGEMENT | 78 |
| 16.1. | Access to Source Data/Document | 78 |
| 16.2. | Confidentiality of Information | 79 |
| 16.3. | Data Quality Assurance | 79 |
| 16.4. | Data Monitoring Committee | 79 |
| 17. C | LINICAL MONITORING | 79 |
| 18. E | THICAL AND REGULATORY ASPECTS | 80 |
| 18.1. | Study-Specific Design Considerations | 80 |
| 18.2. | Investigator Responsibility | 80 |

JJVC CONFIDENTIAL

| 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB) | 80 |
|---|---|
| 18.4. Informed Consent | 81 |
| 18.5. Privacy of Personal Data | 82 |
| 19. STUDY RECORD RETENTION | 83 |
| 20. FINANCIAL CONSIDERATIONS | 84 |
| 21. PUBLICATION | 84 |
| 22. REFERENCES | 84 |
| APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES) | 86 |
| APPENDIX B: PATIENT INSTRUCTION GUIDE | . 107 |
| APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT) | . 108 |
| APPENDIX D: LENS FITTING GUIDE | . 109 |
| APPENDIX E: PRESBYOPIC SYMPTOMS QUESTIONNAIRE | . 113 |
| APPENDIX F: OCULAR DOMINANCE | . 114 |
| APPENDIX G: BINOCULAR OVER REFRACTION | . 115 |
| APPENDIX H: | . 116 |
| , DETERMINATION OF NEAR ADDITION | . 117 |
| , NEAR logMAR VISUAL ACUITY MEASUREMENT PROCEDURE | . 123 |
| , LENS FITTING CHARACTERISTICS | . 126 |
| , SUBJECT REPORTED OCULAR SYMPTOMS | . 132 |
| , DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTI | |
| , BIOMICROSCOPY SCALE | . 140 |
| , KERATOMETRY | . 146 |
| , DISTANCE AND NEAR VISUAL ACUITY EVALUATION | |
| , TORIC FIT EVALUATION | . 153 |
| , DISTANCE LogMAR VISUAL ACUITY MESAUREMENT PROCEDURE | E 158 |
| , VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINAT | |
| PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE | |
| LIST OF FIGURES Figure 1: Study Flowchart | 16 |

## LIST OF TABLES

| Table 1: Test Article |
|----------------------------------------------------------|
| Table 2: Ancillary Supplies |
| Table 3: Time and Events |
| Table 4: Disallowed systemic medications |
| Table 5: Examples of major and minor protocol deviations |
| Table 6: Sample Size Estimates by Study Endpoint |
| Table 7: Historical Data by Endpoint |

### PROTOCOL TITLE, NUMBER, VERSION AND DATE

Protocol Title: Evaluation of the clinical performance of Daily Disposable Silicone Hydrogel

Multifocal Toric Contact Lenses Protocol Number: CR-6542

Version: 4.0

Date: 25 March 2024

#### SPONSOR NAME AND ADDRESS

Johnson & Johnson Vision Care (JJVC) 7500 Centurion Parkway Jacksonville, FL 32256

#### MEDICAL MONITOR



The Medical Monitor must be notified by the clinical institution/site by e-mail, fax, or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

### **AUTHORIZED SIGNATURES**

The signatures below constitutes the approval of this protocol and the attachments and provide the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations<sup>3</sup>, ISO 14155:2020<sup>1</sup>, and the Declaration of Helsinki<sup>2</sup>.

| Author & Study<br>Responsible | | |
|--------------------------------|-------------------------------|------|
| Clinician | See Electronic Signature Page | DATE |
| Clinical Operations<br>Manager | See Electronic Signature Page | |
| | | DATE |
| Biostatistician | See Electronic Signature Page | DATE |
| | | DATE |
| Biostatistics<br>Reviewer | Cao Electronia Cionatura Dago | |
| Keviewei | See Electronic Signature Page | DATE |
| Data Management | See Electronic Signature Page | |
| | | DATE |
| Medical Safety | Car Elastonia Ciamatona Dua | |
| Officer | See Electronic Signature Page | DATE |
| Medical Monitor | See Electronic Signature Page | |
| | | DATE |

| Approver | See Electronic Signature Page | |
|----------|-------------------------------|------|
| | | DATE |

# **CHANGE HISTORY**

| Version | Originator | Description of Change(s) and | Justification | Date |
|---|---|---|---|---|
| | | Section Number(s) Affected | for change | |
| 1.0 | | Original Protocol | N/A | 16 Nov 2023 |
| 2.0 | | Added Medical Monitor as | New | 06 Dec 2023 |
| | | protocol signatory | procedure | |
| 3.0 | | <ul> <li>Updated lens label (Section 6.4)</li> <li>Updated ocular dominance procedure (Appendix F)</li> <li>Updated lighting specifications for VA (Section 7.2)</li> <li>Updated adverse event definitions (Section 13)</li> </ul> | Study lenses<br>being over-<br>labeled | 22 Feb 2024 |
| 4.0 | | <ul> <li>Additional lens build protocol number (Section 6)</li> <li>Added guidance on protocol deviations for missed PRO items (Section 10)</li> </ul> | Several lens<br>lots rebuilt | 25 Mar 2024 |

# **SYNOPSIS**

| Protocol Title | Evaluation of the clinical performance of Daily Disposable |
|---|---|
| | Silicone Hydrogel Multifocal Toric Contact Lenses |
| | JJVC, 7500 Centurion Parkway, Jacksonville, FL 32256 |
| Clinical Phase | Clinical trial phase: Confirmatory (Design Validation Study) |
| | Design control phase: 3 |
| | This study will be registered on ClinicalTrials.gov based on |
| | the following: The purpose of the study is for confirmation of |
| | lens performance, not feasibility. |
| | Investigational Product: JJVC Investigational Multifocal |
| | Toric Contact Lens manufactured in Senofilcon A (C3) |
| | material with UV blocker / HEV filter |
| - | Wear Schedule: The study lenses will be used on a daily |
| | disposable basis. |
| | Replacement Schedule: The study lenses will be replaced each day of wear or if lost or damaged. |
| | Primary Objectives |
| 3 | The primary objectives of this study are to demonstrate that |
| | the investigational multifocal toric contact lens in its final lens |
| | design made on the 3GT platform, meets the validation |
| | requirements with respect to visual acuity (logMAR), |
| | subjective CLUE vision scores, lens fit acceptance, toric fit |
| : | acceptance, and ocular health. |
| | Secondary Objectives |
| , | The secondary objectives of this study are to demonstrate that |
| 1 | the investigational lens meet the users' needs in subjective |
| | CLUE comfort and handling scores and lens fit success. |
| | Although CLUE vision scores are a part of the primary |
| | objectives, an additional secondary objective is to |
| | demonstrate the value proposition of the investigational lens |
| | with respect to subject CLUE vision scores. The value proposition for this product requires a more stringent |
| | threshold, compared to the primary objective, to meet the |
| | user's needs in terms of CLUE vision scores. |
| II 1 | |

| Study Endpoints | Primary Endpoints |
|---|---|
| | 1. Visual Acuity (logMAR)- Distance (4m), |
| | 2. Visual Acuity (logMAR)- Intermediate (64cm) |
| | 3. Visual Acuity (logMAR)- Near (40cm) |
| | 4. CLUE Vision scores |
| | 5. Percentage of eyes with an unacceptable lens fit |
| | 6. Percentage of lens fits with rotation stability within 5 |
| | degrees at 15 minutes after insertion |
| | 7. Percentage of lens fits with absolute rotation error |
| | within 10 degrees at 15 minutes after insertion |
| | 8. Percentage of eyes with Grade 3 or 4 slit lamp findings related to the Test lens |
| | Secondary Endpoints |
| | 1. CLUE Vision scores (with modified criteria) |
| | 2. CLUE Comfort scores |
| | 3. CLUE Handling scores |
| | 4. Lens Fit Success [Number of lenses needed to fit (optimize) the subject's vision] |
| Study Design | This is an open-label, 3-visit, single-arm, dispensing clinical trial. |
| | Approximately 155 subjects will be enrolled with the aim that approximately 140 subjects will complete. At Visit 1, eligible subjects will be fit in the study lenses and dispensed for 7±1 days. Subjects will return for Visit 2 for lens optimization and will be dispensed the optimized pair for 7±1 days. At the follow-up visit (Visit 3), study endpoints will be measured, and the exit evaluation will be performed. |
| | See the flowchart (Figure 1) at the end of the synopsis table |
| | for the schematic of the study visits and procedures of main |
| | observations. |
| Sample Size | Approximately 155 subjects will be enrolled (targeting 93 |
| | myopic and 62 hyperopic subjects with astigmatism) with the |
| | aim of completing 140 subjects (approximately 84 myopes and 56 hyperopes). |
| Study Duration | Each individual subject is expected to attend for 3 study visits |
| | over a period of approximately 2 weeks. The total study |
| | duration from first subject's first visit (FSFV) to last subject's |
| | last visit (LSLV) is expected to be approximately 8 to 12 |
| | weeks. |

| Anticipated Study Population | Healthy male and female volunteers with presbyopia, ametropia (hyperopia or myopia) and astigmatism will be screened as per criteria outlined below. All volunteers will have baseline measurements taken to ensure eligibility. The baseline procedures will occur after informed consent has been obtained. For a detailed list of procedures see the time and events schedule listed below. |
|---|---|
| Eligibility Criteria -<br>Inclusion | Potential subjects must satisfy all of the following criteria to be enrolled in the study: |
| | <ol> <li>Inclusion Criteria following Screening The subject must: <ol> <li>Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.</li> <li>Appear able and willing to adhere to the instructions set forth in this clinical protocol.</li> <li>Be at least 40 and not more than 70 years of age at the time of screening.</li> <li>Own a wearable pair of spectacles if required for their distance vision.</li> <li>Be an adapted soft contact lens wearer in both eyes (i.e. worn lenses for at least 8 hours per day at least two days per week for the past 4 weeks).</li> <li>Be already wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom</li> </ol> </li> </ol> |
| | on the "Presbyopic Symptoms Questionnaire". Inclusion Criteria at Baseline Evaluation: |
| | <ol> <li>7. The subject's distance spherical component of their refraction must be in the range of either -1.25 D to -3.75 D, or +1.25 D to +4.25 D.</li> <li>8. The subject's refractive cylinder must be in the range of -1.00 D to -1.75 D in each eye, with the cylinder axes in the range of either 90° ± 15° or 180° ± 15°.</li> <li>9. The subject's ADD power must be in the range of +0.75 D to +2.50 D in each eye.</li> <li>10. The subject must have best corrected distance visual acuity of 20/20<sup>-3</sup> or better in each eye.</li> </ol> |

# Eligibility Criteria - Exclusion

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

Exclusion Criteria following Screening The subject must not:

- 1. Be currently pregnant or lactating.
- 2. By self-report, have any systemic disease (e.g. Sjögren's Syndrome), allergies, infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g. rheumatoid arthritis), or other diseases, which are known to interfere with contact lens wear and/or participation in the study.
- 3. Use systemic medications that may interfere with contact lens wear or cause blurred vision. See Section 9.1 for additional details regarding excluded systemic medications.
- 4. Currently use ocular medication (with the exception of rewetting drops).
- 5. Have any known hypersensitivity or allergic reaction to single use preservative free rewetting drops or sodium fluorescein.
- 6. Have had any previous, or have any planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, cataract surgery, retinal surgery, etc.).
- 7. Have had previous eyelid injuries, surgeries or procedures which are known to have caused abnormal eyelid position or movement, by self-report.
- 8. Have participated in any contact lens or lens care product clinical trial within 7 days prior to study enrollment.
- 9. Be an employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
- 10. Have a history of amblyopia or strabismus, by self-report.
- 11. Have a history of herpetic keratitis, by self-report.

Exclusion Criteria at Baseline Evaluation The subject must not:

12. Have ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion.

| | 10.77 |
|---|---|
| | 13. Have any Grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal |
| | abnormalities, conjunctival injection) on the FDA scale. |
| Disallowed | Use of any prescription or over-the-counter (OTC) |
| Medications/Interventions | medications that may affect contact lens wear. |
| Wedleations/interventions | See Section 9.1 for details regarding disallowed systemic |
| | medications. |
| Measurements and | logMAR visual acuity charts for distance and near vision. |
| Procedures | Subjective responses for vision, comfort and lens handling |
| | using the CLUE questionnaire, as well as MRD questions. |
| | Lens rotation assessment will be made using a slit lamp |
| | biomicroscope with an adjustable beam orientation and axis |
| | dial, or an eyepiece reticle with axis protractor. |
| Microbiology or Other | None |
| Laboratory Testing | |
| Study Termination | The occurrence of one or more Unanticipated Adverse Device |
| | Effect (UADE), or any SAE where relationship to study agent |
| | cannot be ruled out, may result in stopping the further |
| | dispensing of investigational product. In the event of a UADE |
| | or SAE, the Sponsor Medical Monitor will discuss this with |
| | the Principal Investigator before any further subjects are |
| | enrolled. |
| Ancillary Supplies/ Study- | Non-preserved saline and RevitaLens MPDS. Lens cases for |
| Specific Materials | storage of subject's habitual lenses. Lens vials and caps and |
| | materials for returning worn contact lenses will be supplied to |
| Deing in all Inner stiers to ( ) | sites. |
| Principal Investigator(s) | A full list of Principal Investigators, clinical sites, and |
| and Study | institutions is kept separately from the Study Protocol and is |
| Institution(s)/Site(s) | included in the study Trial Master File. |

Figure 1: Study Flowchart



# COMMONLY USED ABBREVIATIONS, ACRONYMS AND DEFINITIONS OF TERMS

ADD Plus Power Required For Near Use

ADE Adverse Device Effect

AE Adverse Event/Adverse Experience
BCVA Best Corrected Visual Acuity

BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations

CI Confidence Interval or Credible Interval (Bayesian)

CLUE Contact Lens User Experience

COAS Complete Ophthalmic Analysis System

COM Clinical Operations Manager CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

CT Center Thickness

D Diopter

DMC Data Monitoring Committee eCRF Electronic Case Report Form EDC Electronic Data Capture

ETDRS Early Treatment Diabetic Retinopathy Study

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

IB Investigator's Brochure ICF Informed Consent Form

ICH International Conference on Harmonization

IDE Investigational Device Exemption
IEC Independent Ethics Committee
IRB Institutional Review Board

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVC Johnson & Johnson Vision Care, Inc.

LC Limbus Center

logMAR Logarithm of Minimal Angle of Resolution MedDRA<sup>©</sup> Medical Dictionary for Regulatory Activities

MOP Manual of Procedures

MPDS Multi-Purpose Disinfecting Solution

NIH National Institutes of Health

OD Right Eye

OHRP Office for Human Research Protections
OHSR Office for Human Subjects Research

OS Left Eye OU Both Eyes

PD Protocol Deviation

PHI Protected Health Information

PI Principal Investigator
PIG Patient Instruction Guide
PQC Product Quality Complaint
PRO Patient Reported Outcome

QA Quality Assurance QC Quality Control

SAE Serious Adverse Event/Serious Adverse Experience

SAP Statistical Analysis Plan SAS Statistical Analysis System

SD Standard Deviation SLF Slit Lamp Findings

SOP Standard Operating Procedure

UADE Unanticipated Adverse Device Effect

USADE Unanticipated Serious Adverse Device Effect

VA Visual Acuity

#### 1. INTRODUCTION AND BACKGROUND

Johnson & Johnson Vision launched their most recent multifocal contact lens called ACUVUE® OASYS 1-DAY MAX MULTIFOCAL in 2022. The lens is recommended for presbyopes who have up to -0.75 D of refractive cylinder. There is a considerable population of presbyopic patients who have greater than -0.75 D of cylinder, in one or both eyes. Currently there are a limited number of soft toric multifocal lenses available. This study will evaluate the performance of prototype daily disposable multifocal toric lenses with a similar multifocal optics design to ACUVUE® OASYS 1-DAY MAX MULTIFOCAL and manufactured in the same senofilcon A (C3) material with an added high energy visible (HEV) light filter. The performance of the lens will be compared to historical control values.

### 1.1. Name and Descriptions of Investigational Products

Test Article: JJVC Investigational Multifocal Toric Contact Lenses manufactured in Senofilcon A (C3) material with UV blocker / HEV filter Refer to Table 1 in Section 6.1 the protocol.

### 1.2. Intended Use of Investigational Products

The intended use of the Investigational Test lens is for the optical correction of distance and near vision in presbyopic persons with non-diseased eyes who have 0.75D to 1.75D of astigmatism. In this study, the lenses will be used in a population of presbyopes who require +1.25 D to +4.25 D or -1.25 D to -3.75 D of spherical correction, -1.00 D to -1.75 D of cylinder at axes 90°±15° or 180°±15° and ADD powers of +0.75 D to +2.50 D (see Section 3.2).

#### 1.3. Summary of Findings from Nonclinical Studies

All previous pre-clinical findings were deemed satisfactory prior to proceeding with clinical trials on humans. For the most comprehensive nonclinical information regarding JJVC Multifocal Toric Contact Lenses manufactured in senofilcon A material refer to the latest version of the CR-6542 Investigator's Brochure<sup>4</sup>.

#### 1.4. Summary of Known Risks and Benefits to Human Subjects

For the most comprehensive risk and benefit information regarding JJVC Multifocal Toric Contact Lenses manufactured in senofilcon A material refer to the latest version of the CR-6542 Investigator's Brochure<sup>4</sup>.

# 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study

Investigational multifocal toric lenses with similar designs and materials have been evaluated in three prior dispensing clinical studies and one non-dispensing clinical study. A summary of these studies is shown below, and relevant safety information for these studies is included in the CR-6542 Investigator's Brochure<sup>4</sup>.

was a single-arm dispensing evaluation of multifocal toric investigational lenses in a myopic population with against-the-rule astigmatism. Lenses used in this study had a slightly different material formulation than the lenses used in subsequent studies (

and the current CR-6542 study). The study lenses were worn for approximately 2 weeks (with a first follow-up visit after 6-8 days, and second follow-up visit after a further 6-8 days). Forty subjects were enrolled in the study and thirty-seven completed it. No adverse events were reported.

was a single-arm dispensing evaluation of multifocal toric investigational lenses in a hyperopic population with against-the-rule astigmatism. This study tested lenses with an older formulation (same as the one used in same as the one used in later studies). In the 2×3 crossover study design involving 6 visits, subjects wore one of the study lens types for approximately 2 weeks, and the other study lens type for approximately 3 weeks. Thirty-five subjects were enrolled, with 3 screen failures and 3 discontinuations. Of the 29 subjects who completed the study, one was excluded from the Per Protocol Population. One non-significant ocular adverse event which led to the subject being discontinued from the study was determined to be not related to the study lens. Another non-significant ocular adverse event for a subject who completed the study was considered as unlikely related to the test article.

was a single-arm, single-masked dispensing evaluation of multifocal toric investigational lenses with 4 study visits (fitting visit, optimization visit, then follow-up visits after 1 and 2 further weeks of wear). The subjects were required to have distance spherical component of their refraction in the range of either -1.25 D to -3.75 D, or +1.25 D to +3.75 D; and refractive cylinder in the range of -1.00 D to -1.50 D with axes in the range of 90°±30°. Ninety-five subjects were enrolled, of whom 9 were screen failures that were not administered the test article. Of the 86 subjects (48 myopes and 38 hyperopes) who wore the study lens, 2 discontinued the study and 1 was excluded from cohort. As a result, the Per Protocol population was 83 subjects (48 myopes and 35 hyperopes). There were no adverse events reported for the study.

was a bilateral, single-masked, single-visit, non-dispensing crossover study of investigational multifocal toric lenses with cylinder corrections of -1.00 and -1.75 diopters. Lens performance in terms of rotation, initial comfort and lens handling was assessed for participants representing four segments of the population (myopic with with-the-rule astigmatism, myopic with against-the-rule astigmatism, hyperopic with with-the-rule astigmatism, and hyperopic with against-the-rule astigmatism). A total of 102 subjects were enrolled, and all completed the study. No adverse events were reported.

In addition to these multifocal toric studies, a series of studies have been performed on the non-toric multifocal version of the study lens during the development of Acuvue<sup>®</sup> Oasys 1-Day Max Multifocal. Further details of the safety profile of these related lens types are included in the CR-6542 Investigator's Brochure<sup>4</sup>.

### 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

### 2.1. Objectives

### **Primary Objectives**

The primary objectives of this study are to demonstrate that the investigational multifocal toric contact lens in its final lens design made on the 3GT platform, meets the validation requirements with respect to visual acuity (logMAR), subjective CLUE vision scores, lens fit acceptance, toric fit acceptance, and ocular health.

### Secondary Objectives

The secondary objectives of this study are to demonstrate that the investigational lens meet the users' needs in subjective CLUE comfort and handling scores and lens fit success. Although CLUE vision scores are a part of the primary objectives, an additional secondary objective is to demonstrate the value proposition of the investigational lens with respect to subjective CLUE vision scores. The value proposition for this product requires a more stringent threshold, compared to the primary objective, to meet the user's needs in terms of CLUE vision scores.

### 2.2. Endpoints

### 2.2.1. Co-Primary Efficacy Endpoints

### 2.2.1.1. High Luminance High Contrast (HLHC) Binocular logMAR Visual Acuities

Multiple additional assessments of binocular and monocular visual acuity will be made at all three distances (4m, 64cm and, 40cm) during the study, but the binocular measurements taken at the 2-Week follow-up in the optimized lens pair using high contrast letters in bright illuminance conditions will be the primary endpoint. The logMAR visual acuity scores at each position are continuous co-primary endpoints.

- VA will be evaluated for 3 different distances. At distance (4 meters), VA will be assessed using ETDRS Charts; while near (40 cm) and intermediate (64 cm) assessments will be made using reduced Guillon-Poling charts. Additional visual acuity will be measured using high and low contrast charts in bright illuminance conditions.
- Visual acuity will also be measured using high contrast charts in dim illuminance conditions (created by the use of goggles).

  in Appendix H for details regarding the collection of visual acuity (logMAR).

### 2.2.1.2. Subjective Vision CLUE Scores

Subjective vision scores assessed using the Contact Lens User Experience (CLUE<sup>TM</sup>) questionnaire at the 2-Week follow-up in the optimized lens pair will be the co-primary endpoint. The overall vision score is a continuous endpoint.

CLUE is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a

contact-lens wearing population in the US, ages 18-65<sup>9</sup>. Derived CLUE™ scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. A 5-point increase in an average CLUE™ score translates into 10% shift in the distribution of scores for population of soft contact lens wearers.

### 2.2.1.3. Rotational Stability

Rotational stability assessed at least 15 minutes after lens insertion at the dispensing visit (Visit 1) is the co-primary endpoint.

Rotation stability will be assessed for each eye at least 15 minutes after lens insertion at the fitting visit, and also at each follow-up visit. Rotational stability is amount of observed rotational movement of the lens' scribe markings in degrees that occurs while blinking in primary gaze. Rotational stability will be converted into a binary endpoint for the purpose of statistical analyses, where Y=1 if the lens stability with blinks is  $\leq 5^{\circ}$  and Y=0, otherwise.

#### 2.2.1.4. Absolute Rotation Error

Absolute rotation error assessed at least 15 minutes after lens insertion at the dispensing visit (Visit 1) is the co-primary endpoint.

Absolute rotation error is quantified by the absolute value of mis-location of the lens' scribe markings in degrees relative to a vertical reference line. It is measured for each eye at 1, 3 and at least 15 minutes after lens insertion at the fitting visit, and also at each follow-up visit. Absolute rotation error will be converted into a binary endpoint for the purpose of statistical analyses where Y=1 if the absolute toric lens rotation is  $\leq 10^{\circ}$  and Y=0, otherwise.

### 2.2.2. Co-Primary Safety Endpoints

#### 2.2.2.1. Incidence of Unacceptable Lens Fit

The co-primary safety endpoint is the incidence (percentage) of eyes with unacceptable fitting at any time during the study.

Unacceptable lens fit will be assessed at all study visits (scheduled and unscheduled) for each eye. Eyes with multiple unacceptable fitting events and or with multiple criteria met at a given visit will be counted only once. Unacceptable lens fit is a binary response where Y=1 if lens fit is unacceptable and Y=0 otherwise. Lens fit is defined as "unacceptable" if any one of the following criteria is met:

- limbal exposure at primary gaze or with extreme eye movement;
- edge lift;
- excessive movement in primary gaze;
- insufficient movement in all three of the following conditions: primary gaze, up gaze, and push up test.

in Appendix H for additional details regarding lens fit assessments.

## 2.2.2.2. Slit Lamp Findings

The co-primary safety endpoint is the incidence (percentage) of eyes with Grade 3 or higher SLF (including any corneal infiltrates) related to the Test lens.

Slit Lamp Findings (Grade 3 or higher) will be assessed for each subject eye at all study visits (scheduled and unscheduled). SLFs will be evaluated and classified using the FDA Grading scale rating from 0 to 4, where Grade 0 represents the absence of findings and 1 to 4 representing successively worse findings (i.e., Grade 1=trace, Grade 2=mild, Grade 3=moderate and Grade 4=severe). Eyes with multiple SL findings of Grade≥3 at different timepoint during the visit, or with different grade level over time, will be counted only once.

### 2.2.3. Secondary Efficacy Endpoints

- Subjective Handling Scores at the 2-Week follow-up visit will be assessed using the CLUE<sup>TM</sup> questionnaire. The overall mean handling score is a continuous endpoint.
- Subjective Comfort Scores at the 2-Week follow-up visit will be assessed using the CLUE<sup>TM</sup> questionnaire. The overall mean comfort score is a continuous endpoint.
- Subjective Vision Scores at the 2-Week follow-up visit will be assessed using the CLUE<sup>TM</sup> questionnaire. The overall vision score is a continuous endpoint.
- Lens Fit Success is the number of lenses needed to fit (optimize) the subject's vision. Lens fit success is a binary endpoint where, Y=1 if a subject's vision was optimized in four lenses or less, and Y=0, otherwise. The number of lenses needed is determined using lens selection data from both Visit 1 and Visit 2.

### 2.3. Hypotheses

All Co-Primary Efficacy and Safety hypotheses listed below must be statistically significantly demonstrated to satisfy the study objectives.

### 2.3.1. Co-Primary Efficacy Hypotheses

- 1. After approximately 2-weeks of wear, the mean HLHC distance (4 m) visual acuity score of the Test lens will be statistically significantly lower than 0.00 logMAR (equivalent to 20/20 on Snellen Visual Acuity scale).
- 2. After approximately 2-Weeks of wear, the mean HLHC intermediate (64 cm) visual acuity score of the Test lens will be statistically significantly lower than 0.17 logMAR (equivalent to 20/30 on Snellen Visual Acuity scale).
- 3. After approximately 2-Weeks of wear, the mean HLHC near (40 cm) visual acuity score of the Test lens will be statistically significantly lower than 0.17 logMAR (equivalent to 20/30 on Snellen Visual Acuity scale).

- 4. After approximately 2-weeks of wear, the mean CLUE overall *quality of vision* score of the Test lens will be statistically significantly better (greater) than 41 for the <u>myope</u> population.
- 5. After approximately 2-weeks of wear, the mean CLUE overall *quality of vision* score of the Test lens will be statistically significantly better (greater) than 36 for the <a href="https://hyperope.ncbi.nlm.nih.gov/hyperope.
- 6. Following lens settling (at least 15 minutes) at the dispensing visit, the percentage of eyes with Test lens rotational stability with blink  $\leq 5^{\circ}$  will be statistically significantly  $\geq 80\%$ .
- 7. Following lens settling (at least 15 minutes) at the dispensing visit, the percentage of eyes with Test lens absolute rotation  $\leq 10^{\circ}$  will be statistically significantly  $\geq 80\%$ .

### 2.3.2. Co-Primary Safety Hypotheses

- 1. The percentage of eyes with at least one clinically significant slit-lamp finding (Grade 3 or 4) related to the Test lens will be statistically significantly less than 5%.
- 2. The percentage of eyes with an unacceptable Test lens fit will be statistically significantly less than 20%.

### 2.3.3. Secondary Efficacy Hypotheses

A fixed sequence approach will be used to control the type I error. The order of testing secondary hypotheses are as follows:

- 1. After approximately 2-Weeks of wear, the mean CLUE *handling* score of the Test lens will be statistically significantly better (greater) than 46 for the hyperope population.
- 2. After approximately 2-Weeks of wear, the mean CLUE *comfort* score of the Test lens will be statistically significantly better (greater) than 38 for the <u>hyperope</u> population.
- 3. After approximately 2-Weeks of wear, the mean CLUE *handling* score of the Test lens will be statistically significantly better (greater) than 55 for the <u>myope</u> population.
- 4. After approximately 2-Weeks of wear, the mean CLUE overall *quality of vision* score of the Test lens will be statistically significantly better (greater) than 41 for the <a href="https://hyperope.population">hyperope</a> population.
- 5. After approximately 2-Weeks of wear, the mean CLUE *comfort* score of the Test lens will be statistically significantly better (greater) than 51 for the myope population.
- 6. After approximately 2-Weeks of wear, the mean CLUE overall *quality of vision* score of the Test lens will be statistically significantly better (greater) than 46 for the <u>myope</u> population.
- 7. The percentage of subjects who are fit with the optimized lens pair in 4 lenses or less will be statistically significantly better (greater) than 90%.

### 3. TARGETED STUDY POPULATION

#### 3.1. General Characteristics

The population to be studied will consist of adapted contact lens wearers with presbyopia, ametropia (hyperopia or myopia) and astigmatism.

#### 3.2. Inclusion Criteria

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

Inclusion Criteria following Screening The subject must:

- 1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
- 2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
- 3. Be at least 40 and not more than 70 years of age at the time of screening.
- 4. Own a wearable pair of spectacles if required for their distance vision.
- 5. Be an adapted soft contact lens wearer in both eyes (i.e. worn lenses for at least 8 hours per day at least two days per week for the past 4 weeks).
- 6. Be already wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".

Inclusion Criteria at Baseline Evaluation

- 7. The subject's distance spherical component of their refraction must be in the range of either -1.25 D to -3.75 D, or +1.25 D to +4.25 D.
- 8. The subject's refractive cylinder must be in the range of -1.00 D to -1.75 D in each eye, with the cylinder axes in the range of either 90°±15° or 180°±15°.
- 9. The subject's ADD power must be in the range of +0.75 D to +2.50 D in each eye.
- 10. The subject must have best corrected distance visual acuity of 20/20<sup>-3</sup> or better in each eye.

### 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

Exclusion Criteria following Screening The subject must not:

- 1. Be currently pregnant or lactating.
- 2. By self-report, have any systemic disease (e.g. Sjögren's Syndrome), allergies, infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g. rheumatoid arthritis), or other diseases, which are known to interfere with contact lens wear and/or participation in the study.

- 3. Use systemic medications that may interfere with contact lens wear or cause blurred vision. See Section 9.1 for additional details regarding excluded systemic medications.
- 4. Currently use ocular medication (with the exception of rewetting drops).
- 5. Have any known hypersensitivity or allergic reaction to single use preservative free rewetting drops or sodium fluorescein.
- 6. Have had any previous, or have any planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, cataract surgery, retinal surgery, etc.).
- 7. Have had previous eyelid injuries, surgeries or procedures which are known to have caused abnormal eyelid position or movement, by self-report.
- 8. Have participated in any contact lens or lens care product clinical trial within 7 days prior to study enrollment.
- 9. Be an employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
- 10. Have a history of amblyopia or strabismus, by self-report.
- 11. Have a history of herpetic keratitis, by self-report.

Exclusion Criteria at Baseline Evaluation The subject must not:

- 12. Have ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion.
- 13. Have any Grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA scale.

### 3.4. Enrollment Strategy

Study subjects will be recruited from the Institution/clinical site's subject database and/or utilizing Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved materials.

In order to enroll a study population which is reasonably representative of the presbyopic contact lens market, the enrolment targets have been designed based on a 60:40 ratio between myopes and hyperopes for the total study population. Individual sites will also be asked to try to enroll myopes and hyperopes according to this ratio, when possible.

In order to ensure that the performance of study lenses with Low, Mid and High near addition power are tested in this study, study sites will be asked to try, when possible, to enroll at least one myopic and one hyperopic subject that have a near ADD requirement in each of these ranges ( $\pm 0.75$  to  $\pm 1.25$  D,  $\pm 1.50$  to  $\pm 1.75$  D, and  $\pm 2.00$  to  $\pm 2.50$  D).

#### 4. STUDY DESIGN AND RATIONALE

### 4.1. Description of Study Design

This is an open-label, single-arm, 3-visit, dispensing clinical trial. Approximately 155 subjects (93 myopes and 62 hyperopes) will be enrolled into the study with the aim of completing approximately 140 subjects (84 myopes and 56 hyperopes).

The study begins with an initial visit, Visit 1 (Day 0), then if a subject is found to meet all eligibility criteria, they will be fit with the study lens in both eyes. Otherwise, the subject will be deemed ineligible and classified as a screen failure and exited from the study.

If a subject is dispensed lenses at the initial visit, then two additional visits will be conducted. Visit 2 will be conducted  $7\pm1$  days after Visit 1, where subjects will undergo lens optimization, if needed. Subjects will be dispensed the optimized pair for  $7\pm1$  days and return for Visit 3. Study endpoints will be measured, and the subject will be exited from the study.

Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day between visits. Lost or damaged lenses may be replaced when necessary. Unscheduled visits may be conducted, if necessary.

### 4.2. Study Design Rationale

The objective of this study is to demonstrate that the investigational lens, in its final design, meets criteria for visual acuity (logMAR), CLUE scores, lens fit attributes, and ocular health compared to predefined thresholds specified in the Customer Requirements Document (Therefore, a single-arm study was chosen as the appropriate design to test co-primary efficacy and safety hypotheses.

### 4.3. Enrollment Target and Study Duration

Approximately 155 subjects will be enrolled with the aim that approximately 140 subjects will complete. The study will be conducted at up to 16 clinical sites. Approximately 93 myopic subjects with astigmatism will be enrolled, with the aim that at least 84 will complete the study. Approximately 62 hyperopic subjects with astigmatism will be enrolled, with the aim that at least 56 will complete the study. Each individual subject is expected to attend for 3 study visits over a period of approximately 2Weeks. The total study duration from first subject's first visit (FSFV) to last subject's last visit (LSLV) is expected to be approximately 8 to 12 weeks.

### 5. TEST ARTICLE ALLOCATION AND MASKING

### 5.1. Test Article Allocation

This is a single-arm study. All eligible subjects will be dispensed the study lens in a bilateral fashion.

### 5.2. Masking

This is considered an open-label trial as there is only one type of study lens. The subjects will be aware of the type of contact lens to be dispensed in this study, but will not be aware of the specifics of the lens design, beyond that the lenses are intended to correct for their distance and near vision. Neither investigators nor clinical site personnel involved in the data collection will be masked as to the identity of the investigational product.

### 5.3. Procedures for Maintaining and Breaking the Masking

Not applicable.

### 6. STUDY INTERVENTION

## 6.1. Identity of Test Articles

The following investigational contact lens will be used in this study:

Table 1: Test Article

| | Test Lens |
|--------------------------------------|---------------------------------------|
| Name | JJVC Investigational Multifocal Toric |
| | Contact Lenses manufactured in |
| | Senofilcon A (C3) material with UV |
| | blocker / HEV filter |
| Design | AMT series |
| Manufacturer | JJVC |
| Packaging Form (vial, blister, etc.) | Blister |
| Lens Material | senofilcon A(C3) with chromophore |
| Nominal Base Curve | 8.5 |
| Nominal Diameter | 14.3 |
| Nominal Distance Powers (D) | -1.00 to -4.00 in 0.25D steps, |
| | +1.00 to +4.50 in 0.25D steps |
| Nominal Cylinder Powers (D) | -1.00 |
| Cylinder axes (°) | 10, 80, 90, 100, 170, 180 |
| Nominal ADD Power (D) | Low, Mid, High |
| Fiducial marks | 6 and 12 o'clock fiducial lines |
| Water Content | 38% |
| Oxygen Permeability (Dk) | 122.0 |
| Wear Schedule in Current Study | Daily Disposable |
| Replacement Frequency | Daily |

Each subject will wear approximately 32 lenses for the average 14 day dispensing period, including the 2 lenses provided at Visit 1, and 2 new lenses provided at Visit 2. Additional lenses may be used as needed for power modifications and replacements.

### 6.2. Ancillary Supplies/Products

The following solutions will be used in this study:

Table 2: Ancillary Supplies

| | Single-Use Preservative-Free Rewetting Solutions (any of these three options may be supplied) | | Multipurpose<br>Solution | |
|---|---|---|---|---|
| Solution<br>Name /<br>Description | Eye-Cept <sup>®</sup><br>Rewetting<br>Drops | ScleralFil®<br>Preservative Free<br>Saline Solution | LacriPure<br>Saline<br>Solution | Acuvue <sup>TM</sup> RevitaLens Multi-Purpose Disinfecting Solution (MPDS) |
| Manufacturer | Optics<br>Laboratory | Bausch + Lomb | Menicon | Johnson &<br>Johnson Vision |
| Preservative | Non-Preserved | Non-Preserved | Non-<br>Preserved | alexidine<br>dihydrochloride<br>0.00016% and<br>polyquaternium-1<br>0.0003% |

Stopwatches will be provided to research sites to help with managing the timing of toric fit assessments and lens settling.

Contact lens cases will be provided for storage of a subject's habitual contact lenses that they wish to keep for reuse.

Note: RevitaLens MPDS is provided for the purpose of temporary storage of a subject's habitual lenses that they remove at Visit 1. It may also be used for the storage of study lenses that need to be returned to the sponsor (ie. lenses associated with a Product Quality Complaint or Adverse Event). RevitaLens solution will not be provided to the subject for use at home with the study lenses, since the study lenses are daily disposable.

#### 6.3. Administration of Test Articles

Test article will be dispensed to subjects meeting all eligibility requirements, including any dispensing requirements set forth in this clinical protocol. Subjects will be dispensed an adequate supply of test articles to complete the study. Test articles which are lost or damaged may be replaced at the discretion of the Investigator.

### 6.4. Packaging and Labeling

The Test article will be packaged in blisters as the primary packaging with an investigational lens label. The test article will be in plastic bags as the secondary packaging form. The sample study label is shown below:

Primary Packaging



Secondary Packaging



#### 6.5. Storage Conditions

Test articles will be maintained at ambient temperatures at the clinical site. Test articles must be kept under secure conditions.

#### 6.6. Collection and Storage of Samples

When possible, any lens or test article associated with an Adverse Event and/or a Product Quality Complaint must be retained and stored in a glass vial with saline or MPDS solution pending directions from the sponsor for potential return to JJVC.

#### 6.7. Accountability of Test Articles

JJVC will provide the Investigator with sufficient quantities of study articles and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test articles must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted for. This includes:

- 1. What was dispensed for the subject for trial fitting, to wear out of the office, or issued for the subject to replace appropriately between visits.
- 2. What was returned to the Investigator unused, including expired or malfunctioning product.
- 3. The number and reason for unplanned replacements.

The Investigator will collect all unused test articles from the subjects at the end of the subject's participation. Subject returned unused test articles must be separated from the clinical study inventory of un-dispensed test articles and must be labeled with the subject number and date of return. Following final reconciliation of test articles by the monitor, the Investigator or monitor will return all unused test articles to JJVC.

If there is a discrepancy between the shipment documents and the contents, contact the study monitor immediately.

#### 7. STUDY EVALUATIONS

#### 7.1. Time and Event Schedule

Table 3: Time and Events

| Visit Information | Visit 1 | Visit 2 | Visit 3 |
|---|---|---|---|
| | Screening, | Treatment 1 Follow- | Treatment 1 Follow- |
| | Baseline, Treatment | up 1 | up 2 |
| | 1 | | |
| Time Point | Day 0 | 7 ± 1 days after Visit | $7 \pm 1$ days after Visit |
| | | 1 | 2 |
| Estimated Visit Duration | 2.5 hours | 1.5 hours | 1.0 hours |
| Statement of Informed Consent | X | | |
| Demographics | X | | |
| Medical History/Concomitant | X | | |
| Medications/Review | Λ | | |
| AE/Concomitant Med Review | | X | X |
| Habitual Contact Lens Information & | X | | |
| Wear Schedule | Λ | | |
| Contact Lens History | X | | |
| Habitual Lens Wear Time | X | | |
| Study Lens Wear Time | | X | X |
| Compliance | | X | X |
| Presbyopic Symptoms Questionnaire | X | | |
| Screening Inclusion/Exclusion | X | | |
| Criteria | Λ | | |

| Visit Information | Visit 1<br>Screening,<br>Baseline, Treatment | Visit 2<br>Treatment 1 Follow-<br>up 1 | Visit 3<br>Treatment 1 Follow-<br>up 2 |
|---|---|---|---|
| Time Point | Day 0 | 7 ± 1 days after Visit<br>1 | 7 ± 1 days after Visit<br>2 |
| Estimated Visit Duration | 2.5 hours | 1.5 hours | 1.0 hours |
| Patient Reported Outcomes | X | X | X |
| Ocular Symptoms | X | X | X |
| Subjective Acceptance | | X | X |
| Entrance distance and near Visual | X | X | X |
| Acuity | Λ | Λ | Λ |
| Lens Removal | X | X | X |
| Keratometry | X | | |
| Subjective Sphero-Cylindrical<br>Refraction | X | | |
| Near ADD Determination | X | | |
| Ocular Dominance | X | | |
| ADD Refinement | X | | |
| Near Visual Acuity | X | | |
| Slit Lamp Biomicroscopy | X | X | X |
| Baseline Inclusion/ Exclusion | X | | |
| First choice lens power | X | | |
| Lens Selection | XOO | 00 | |
| Right Lens Insertion | XOO | | |
| Right Lens 1 Minute and 3 Minute<br>Rotation | XOO | | |
| Left Lens Insertion | XOO | | |
| Left Lens 1 Minute and 3 Minute | | | |
| Rotation | XOO | | |
| Lens Settling | XOO | 00 | |
| Toric Fit Evaluation | XOO | XOO | X |
| Subjective Lens Fit Assessment | XOO | XOO | X |
| Visual Satisfaction | XOO | 00 | |
| Study Lens Distance and Near Visual<br>Acuity | XOO | 00 | |
| Over Refraction and Visual Acuity | XOO | XOO | X |
| Lens Power Modification (if required) | X | X | 71 |
| Additional Lens Power Modification<br>(if required) | | X | |
| Collect unworn study lenses (if | | X | X |
| applicable) | | | v |
| Visual Performance | | X | X |
| Insert new pair of lenses Exit Snellen Distance and Near Visual | X | X | |
| Acuity | | | |
| Dispensing Criteria | X | X | |
| Dispensing | X | X | |
| Subject Instructions | X | X | |
| Schedule Follow-Up | X | X | |
| Final Evaluation | | | X |

Note: O denotes Optional items performed if required based on results

# 7.2. Detailed Study Procedures

### VISIT 1

Subjects must report to the visit wearing their habitual contact lenses to accurately assess baseline PRO (CLUE and MRD) performance. If the subject is not wearing their lenses they must be rescheduled.

| | Visit 1: Screening | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.1 | Statement of<br>Informed Consent | Each subject must read, understand, and sign the Statement of Informed Consent before being enrolled into the study. The Principal Investigator or his/her designee conducting the informed consent discussion must also sign the consent form. | |
| | | <u>Note</u> : The subject must be provided a signed copy of this document. | |
| 1.2 | Demographics | Record the subject's year of birth, age, sex, race and ethnicity. | |
| 1.3 | Medical History and<br>Concomitant<br>Medications | Questions regarding the subject's medical history and concomitant medications. | |
| 1.4 | Habitual Contact<br>Lens Information | Questions regarding the subject's habitual lens type and parameters. | |
| 1.5 | Habitual Contact<br>Lens Wear Schedule | Record the duration of wearing this contact lens type and power (number of years and months). During the past four weeks, what is the minimum number of days per week that the subject has worn their lenses for at least 8 hours. | |
| 1.6 | Contact Lens History | Record the subject's correction type (i.e. monovision, multifocal, sphere with readers, etc.). | |
| 1.7 | Wear time and<br>Comfortable Wear<br>time with Habitual<br>lenses | Record the subject's wear time and comfortable wear time with their habitual contact lenses. | |
| 1.8 | Presbyopic<br>Symptoms<br>Questionnaire | Subjects will be asked if they are wearing a presbyopic correction and whether they are experiencing any of five common symptoms of presbyopia. | Appendix<br>E |
| 1.9 | Eligibility after<br>Screening | All responses to Screening Inclusion Criteria questions must be answered "yes" and all | |

| | Visit 1: Screening | |
|---|---|---|
| Step | Procedure | Details |
| | | responses to Exclusion Criteria must be |
| | | answered "no" for the subject to be |
| | | considered eligible. |
| | | If subject is deemed to be ineligible after screening, proceed to Final Evaluation and complete Subject Disposition. Refraction and Biomicroscopy forms are not required. |

| | Visit 1: Baseline | |
|---|---|---|
| Step | Procedure | Details |
| 1.10 | Baseline PRO<br>(CLUE and MRD)<br>Questionnaires | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms |
| | | of their habitual lenses using the PRO (CLUE and MRD) questions. |
| 1.11 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| 1.12 | Entrance Distance<br>and Near Visual<br>Acuity | Record the distance and near Snellen visual acuity (OD, OS, OU) to the nearest letter with the subject's habitual contact lenses in place. For near measurements use the ETDRS 2000 Series Chart 1 or 2. If the subject habitually wears reading glasses over their contact lenses, these may be worn for near acuity. |
| 1.13 | Lens Removal | Have the subject remove their habitual lenses and store in an approved storage solution. RevitaLens MPDS is supplied for the study, but an alternative MPDS may be used. |
| 1.14 | Keratometry / SimK | Keratometry/SimK will be performed OD and OS and the steep and flat dioptric power and corresponding meridians recorded. |
| 1.15 | Subjective Sphero-<br>cylindrical<br>Refraction | An optimal, binocular balanced distance sphero-cylindrical refraction will be performed. Record the refraction and distance visual acuity (OD, OS, OU) to the nearest letter. Note: Best distance visual acuity with sphero-cylindrical refraction must be at least 20/20 <sup>3</sup> in each eye for the subject to be eligible in the study. |

| | Visit 1: Baseline | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.16 | Near ADD | The near reading addition will be determined | |
| | Determination | using the binocular crossed cylinder | |
| | | technique (BCC) at 40 cm | |
| 1.17 | Ocular Dominance | Determine the distance ocular dominance | Appendix |
| | | with the best distance correction in place | F |
| | | using a +1.00-blur test. If the amount of blur | |
| | | appears the same for the two eyes, then try a | |
| | | +1.50 D lens. | |
| | | If the results are equivocal use the sighting | |
| | | dominance test to determine the dominant eye | |
| | | used for the study. | |
| 1.18 | ADD Refinement | Place the BCC result in the trial frame and | |
| | | refine the near prescription with trial lenses | |
| 1.10 | 37 77 1 A 14 | (or flippers) under binocular conditions. | |
| 1.19 | Near Visual Acuity | Using the ETDRS 2000 Series Chart 1 or 2 | |
| | | near card placed at 40 cm. Record the near | |
| 1.20 | D:: | visual acuity (OD, OS, OU). | |
| 1.20 | Biomicroscopy | FDA Slit Lamp Classification Scale will be | |
| | | used to grade the findings and determine eligibility. | |
| | | engionity. | |
| | | If any of these slit lamp findings are Grade 3 | |
| | | or higher, the subject will be discontinued. If | |
| | | discontinued a final examination must be | |
| | | completed. | |
| | | If the clearance of the fluorescein needs to be | |
| | | expedited, preservative-free saline may be | |
| | | instilled. | |
| 1.21 | Eligibility after | All responses to Inclusion Criteria questions | |
| | Baseline | must be answered "yes" and all responses to | |
| | | Exclusion Criteria questions must be | |
| | | answered "no" for the subject to be | |
| | | considered eligible. | |
| | | If subject is deemed to be ineligible after | |
| | | baseline, proceed to Final Evaluation and | |
| | | complete all forms. | |

| | Visit 1: Treatment 1 Lens Fitting | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.22 | First choice lens | Record the first choice lens' sphere power, | Appendix |
| | powers | cylinder power, axis and add for each eye | D |

| Visit 1: Treatment 1 Lens Fitting | | | | |
|---|---|---|--|--|
| Step | Procedure | Details | | |
| | | based on the refraction and fitting guide, by considering: | | |
| | | Lens powers available in the study. | | |
| | | Adjustment of sphere power for | | |
| | | vertex distance (if needed) | | |
| | | Adjustment of sphere power to | | |
| | | compensate for any under-correction | | |
| | | of cylinder by the available study lens | | |
| | | (at the investigator's discretion) | | |
| | | Closest available axis. If refractive | | |
| | | cylinder axis is 5 degrees away from | | |
| | | two available lens axes, either may be | | |
| | | chosen at the investigator's discretion | | |
| | | The final near add which was | | |
| | | determined and the dominant eye | | |
| 1.23 | Lens Selection | Select the lens power and axis based on the | | |
| | | first choice lens powers determined in the | | |
| | | previous step. Record the test lens | | |
| 1.24 | Dight I and Industion | parameters (power and lot number). | | |
| 1.24 | Right Lens Insertion | Subjects will insert the right lens themselves. If the lens is uncomfortable, inspect for | | |
| | | damage and remove, reinsert or replace as | | |
| | | necessary. | | |
| | | necessary. | | |
| | | Damaged lenses will be stored in a labeled | | |
| | | vial with saline for shipment back to the | | |
| | | Sponsor. Complete the Product Quality | | |
| | | Complaint form. | | |
| 1.25 | Timed Settling for | The investigator will start a stopwatch as | | |
| | Right Lens | soon as the right lens is inserted. | | |
| | | Note: All lenses in this study have toric | | |
| | | orientation marks at the 6 and 12 o'clock | | |
| | | positions. Rotation measurements are | | |
| | | made relative to a vertical reference line. | | |
| | | Direction of rotation is recorded as base | | |
| | | nasal or base temporal. | | |
| | | At one (1) minute after insertion, record the | | |
| | | rotational position to the nearest degree. | | |
| | | At three (3) minutes after insertion, record the | | |
| | | rotational position to the nearest degree. | | |
| | , | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|--|
| Step | Procedure | Details | |
| 1.26 | Left Lens Insertion | Subjects will insert the left lens themselves. If<br>the lens is uncomfortable, inspect for damage<br>and remove, reinsert or replace as necessary. | |
| | | Damaged lenses will be stored in a labeled vial with saline for shipment back to the Sponsor. Complete the Product Quality Complaint form. | |
| 1.27 | Timed Settling for<br>Left Lens | The investigator will start a stopwatch as soon as the left lens is inserted. | |
| | | Note: All lenses in this study have toric orientation marks at the 6 and 12 o'clock positions. Rotation measurements are made relative to a vertical reference line. Direction of rotation is recorded as base nasal or base temporal. | |
| | | At one (1) minute after insertion, record the rotational position to the nearest degree. | |
| | | At three (3) minutes after insertion, record the rotational position to the nearest degree. | |
| 1.28 | Lens Settling | Allow the study lenses to settle for a minimum of 15 minutes from the time of last lens insertion. | |
| 1.29 | Toric Fit Evaluation | Record: • The rotational position to the nearest degree • Lens stability with blink • Toric fit acceptable or unacceptable Toric lens fit will be unacceptable if lenses rotated more than 30 degrees, or lens stability is worse than 5 degrees movement with blink. If toric fit is unacceptable for either eye, the subject will be discontinued from the study. Remove and discard the | |
| 1.30 | Lens Fit Assessment | lenses, then proceed to Final Evaluation. Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). | |
| | | J T P | |

| | Visit 1: Treatment 1 Lens Fitting | | |
|---|---|---|---|
| Step | Procedure | Details | |
| | | Lens fit will be unacceptable if any of the | |
| | | following is observed: | |
| | | <ul> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> <li>presence of edge lift</li> <li>presence of excessive movement with blink in primary gaze</li> <li>presence of insufficient movement in all three movement categories (primary gaze, upgaze, and push-up test).</li> </ul> | |
| | | If lens fit is unacceptable for either eye, the subject will be discontinued from the study. Remove and discard the lenses, then proceed to Final Evaluation. | |
| 1.31 | Determine Visual<br>Satisfaction | Determine if the subject's vision is acceptable with the lenses. Allow the subject to look down a hallway or out of a window for distance vision assessments, and for them to read a book, magazine or similar for near vision. | |
| 1.32 | Study Lens Distance<br>and Near Visual<br>Acuity | Record the distance and near Snellen visual acuity (OD, OS, OU) to the nearest letter with the study contact lenses in place. For near measurements use the ETDRS 2000 Series Chart 1 or 2. | |
| 1.33 | Distance Over-<br>Refraction and<br>Distance Visual<br>Acuity | Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. | |
| 1.34 | Lens Power<br>Modification (if<br>applicable) | If the subject reports unsatisfactory vision, or is unable to obtain 20/30 distance visual acuity OU with the lenses, then a modification must be attempted. If the subject reports satisfactory vision with the lenses a modification is not required; however it may be made at the Investigators discretion based | Appendix<br>D |

| | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| | | upon their findings on the measured visual acuity and/or over- refraction. Note: switching to a non-multifocal lens per Step 3 of the Fitting Guide is not an available option in this study. |
| | | Select the reason(s) for lens change (select all that apply): • The settled lens rotation is such that one of the other available lens cylinder axes would be better (use LARS rule to determine the replacement lens cylinder axis) • Power Modification needed • Unsatisfactory Vision • Other (specify reason) |
| | | If one or both lenses are modified, repeat steps <b>1.23 through 1.34</b> for one or both eyes as appropriate. A maximum of <i>two</i> lens modifications are allowed. |
| 1.35 | Exit Distance and<br>Near Visual Acuity | Record the distance and near Snellen visual acuity (OD, OS, OU) to the nearest letter with the study contact lenses in place. For near measurements use the ETDRS 2000 Series Chart 1 or 2. |
| 1.36 | Dispensing<br>Criteria | <ul> <li>The lenses may be dispensed for 6-8 days, if the following criteria are met:</li> <li>Distance Snellen acuity equal to or better than 20/30 OU</li> <li>Subject must indicate that the vision is acceptable.</li> <li>Subject must indicate that the comfort of the lenses is acceptable.</li> <li>Lenses must have an acceptable toric and general lens fit.</li> </ul> |
| 1.37 | Dispensing | Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No spare lenses will be dispensed. |
| 1.38 | Subject Instructions | <ul> <li>Instruct the Subject on the following:</li> <li>The lenses will be worn on a daily disposable wear basis.</li> </ul> |

| | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details Details |
| Step | Procedure | <ul> <li>Instruct the subject to bring back all unworn study lenses.</li> <li>Instruct the subject no cleaning or disinfecting solutions will be used for this lens type.</li> <li>If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day between visits. One missed day of lens wear between visits is acceptable.</li> <li>Subjects will be instructed to wear study lenses to the next visit. It is not required that they have worn lenses for 6 hours on the day of the visit.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>A patient instruction booklet will be provided.</li> <li>Note: In the event a lens is lost or damaged, the subject may return to the investigator site for a replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in a labeled vial with saline or MPDS solution and returned to the Sponsor.</li> </ul> |
| 1.39 | Schedule<br>Follow-up | The subject will be scheduled to return for their follow-up appointment in 7±1 days. |

VISIT 2

The subjects must present to Visit 2 wearing the study lenses.

| | Visit 2: Treatment 1 Follow-Up 1 | |
|---|---|---|
| Step | Procedure | Details |
| 2.1 | Adverse Events and | Review any changes to the subject's medical |
| | Concomitant | history or concomitant medications from the |
| | Medications Review | previous study visit. Record any changes, |
| | | and any adverse events. |
| 2.2 | Wear time and | Record the average wearing time and |
| | Comfortable Wear | comfortable wearing time with the study |
| | time (Study Lenses) | lenses. |
| 2.3 | Compliance | Confirm compliance with the prescribed |
| 2.0 | Compilation | wear schedule. |
| 2.4 | Collect unworn study | Any remaining unworn study lenses will be |
| | lenses (if applicable) | collected from the subject. |
| 2.5 | PRO (CLUE and | The subject will respond to the Follow-Up |
| | MRD) Questionnaires | PRO (CLUE and MRD) Questionnaires. |
| 2.6 | Subject Reported | Subjects will respond to a verbal open-ended |
| | Ocular Symptoms | symptoms questionnaire. |
| 2.7 | Subjective Acceptance | Record whether the subject's distance and |
| | , , | near vision with the lenses is acceptable. |
| 2.8 | Entrance Distance and | Record the distance and near Snellen visual |
| | Near Visual Acuity | acuity (OD, OS, OU) to the nearest letter with |
| | | the study contact lenses in place. |
| | | For near measurements use the ETDRS |
| | | 2000 Series Chart 1 or 2. |
| 2.9 | Distance Over- | Perform a distance over-refraction OD and |
| , | Refraction and | OS using loose lenses outside of the |
| | Distance Visual Acuity | phoropter under ambient room illumination. |
| | Distance Visual Fredity | The distance over-refraction may also be |
| | | refined under binocular conditions. |
| | | Record the results. The results of the |
| | | distance over-refraction may also be checked |
| | | for the impact on near vision under |
| | | monocular and/or binocular conditions. |
| 2.10 | Toric Fit Evaluation | Record: |
| | | The rotational position to the nearest |
| | | degree |
| | | 1 |
| | | Lens stability with blink The following the state of the state o |
| | | Toric fit acceptable or unacceptable |
| | | Toric lens fit will be unacceptable if lenses |

| | Visit 2: Treatment 1 Follow-Up 1 | |
|---|---|---|
| Step | Procedure | Details |
| | | rotated more than 30 degrees, or lens stability is worse than 5 degrees movement with blink. If toric fit is unacceptable for either eye, the subject will be discontinued from the study. Remove and discard the |
| | | lenses, then proceed to Final Evaluation. |
| 2.11 | Lens Fit Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). Lens fit will be unacceptable if any of the following is observed: |
| | | <ul> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> <li>presence of edge lift</li> <li>presence of excessive movement with blink in primary gaze</li> <li>presence of insufficient movement in all three movement categories (primary gaze, upgaze, and push-up test).</li> </ul> |
| | | If lens fit is unacceptable for either eye, the subject will be discontinued from the study. Remove and discard the lenses, then proceed to Final Evaluation. |
| 2.12 | Lens Power<br>Modification (if<br>required) | If the subject's vision is unacceptable for at least one distance or the Investigator determines that the visual acuity or overrefraction are not acceptable then a lens modification must be made. If modifications are not needed, proceed to step 2.22. Up to two attempts at changes are permitted, if necessary, in order to achieve an acceptable distance and near binocular performance for the subject. |
| | | Select the reason(s) for lens change (select all that apply): • The settled lens rotation is such that one of the other available lens cylinder axes would |

| | Visit 2: Treatment 1 Follow-Up 1 | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 3.00 | 22000 | be better (use LARS rule to determine the replacement lens cylinder axis) • Power Modification needed • Unsatisfactory Vision • Other (specify reason) | |
| | | Note: switching to a non-multifocal lens per<br>Step 3 of the Fitting Guide is not an<br>available option in this study. | |
| 2.13 | Lens Selection (if required) | Select the lens power, based on the Fitting Guide for each eye needing optimization. Record the test lens parameters (power and lot number). | Appendix<br>D |
| 2.14 | Lens Insertion (if required) | Subjects will insert the lens themselves. If the lens is uncomfortable, inspect for damage and remove, reinsert or replace as necessary. Damaged lenses will be stored in labeled vial with saline solution, and clearly differentiated from the other worn lenses that will be shipped back to the Sponsor. Complete the Product Quality Complaint form. | |
| 2.15 | Lens Settling (if required) | Allow the study lenses to settle for a minimum of 15 minutes from the time of last lens insertion. | |
| 2.16 | Toric Fit Evaluation (if required) | Record: • The rotational position to the nearest degree • Lens stability with blink • Toric fit acceptable or unacceptable Toric lens fit will be unacceptable if lenses rotated more than 30 degrees, or lens stability is worse than 5 degrees movement with blink. If toric fit is unacceptable for either eye, the subject will be discontinued from the study. Remove and discard the lenses, then proceed to Final Evaluation. | |

| | Visit 2: Treatment 1 Follow-Up 1 | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 2.17 | Lens Fit Assessment (if required) | | |
| | | Lens fit will be unacceptable if any of the following is observed: • presence of limbal exposure (appearance of clear cornea) in any gaze • presence of edge lift • presence of excessive movement with blink in primary gaze • presence of insufficient movement in all three movement categories (primary gaze, upgaze, and push-up test). | |
| | | If lens fit is unacceptable for either eye, the subject will be discontinued from the study. Remove and discard the lenses, then proceed to Final Evaluation. | |
| 2.18 | Determine Visual<br>Satisfaction (if<br>required) | Determine if the subject's vision is acceptable with the lenses. Allow the subject to look down a hallway or out of a window for distance vision assessments, and for them to read a book, magazine or similar for near vision. | |
| 2.19 | Study Lens Distance<br>and Near Visual<br>Acuity (if required) | Record the distance and near Snellen visual acuity (OD, OS, OU) to the nearest letter with the study contact lenses in place. For near measurements use the ETDRS 2000 Series Chart 1 or 2. | |
| 2.20 | Distance Over-<br>Refraction and<br>Distance Visual Acuity<br>(if required) | Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. | |
| 2.21 | Additional Lens Power<br>Optimization (if<br>required) | If the subject reports unsatisfactory vision, or is unable to obtain 20/30 distance visual acuity OU with the lenses, then a modification must be attempted. If the | Appendix<br>D |

| | Visit 2: Treatment 1 Follow-Up 1 | |
|---|---|---|
| Step | Procedure | Details |
| | | subject reports satisfactory vision with the lenses a modification is not required however may at the Investigators discretion based upon their findings on the measured visual acuity and/or over- refraction. Note: switching to a non-multifocal lens per Step 3 of the Fitting Guide is not an available option in this study. |
| | | Select the reason(s) for lens change (select all that apply): • The settled lens rotation is such that one of the other available lens cylinder axis would be better (use LARS rule to determine the replacement lens cylinder axis) • Power Modification needed • Unsatisfactory Vision • Other (specify reason) If one or both lenses are modified, repeat |
| | | steps <b>2.13 through 2.20</b> for one or both eyes as appropriate. |
| 2.22 | Lens Removal | Have the subject remove the study lenses. Temporarily store the worn lenses until Biomicroscopy has been completed. If no adverse event or PQC was recorded, the worn lenses may be discarded. |
| 2.23 | Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings. If the clearance of the fluorescein needs to be expedited, preservative-free saline may be instilled. If the subject has a Grade 3 or worse slit lamp finding, it will be recorded as an Adverse Event and the subject will be monitored as per the guidelines given in section 13. |
| 2.24 | Insertion of Study<br>Lenses | Provide the subject with a <b>NEW PAIR</b> of lenses that match the power of the lenses that were removed in step 2.22 above. |
| 2.25 | Exit Distance and<br>Near Visual Acuity | Record the distance and near Snellen visual acuity (OD, OS, OU) to the nearest letter with the study contact lenses in place. |

| | Visit 2: Treatment 1 Follow-Up 1 | |
|---|---|---|
| Step | Procedure | Details |
| | | For near measurements use the ETDRS |
| | | 2000 Series Chart 1 or 2. |
| 2.26 | Dispensing<br>Criteria | The lenses may be dispensed for 6-8 days, if the following criteria are met: • Distance Snellen acuity equal to or better than 20/30 OU • Subject must indicate that the vision is acceptable. • Subject must indicate that the comfort of the lenses is acceptable. • Lenses must have an acceptable toric and general lens fit. |
| 2.27 | Dispensing | Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No spare lenses will be dispensed. |
| 2.28 | Subject Instructions | <ul> <li>Instruct the Subject on the following:</li> <li>The lenses will be worn on a daily disposable wear basis.</li> <li>Instruct the subject to bring back all unworn study lenses.</li> <li>Instruct the subject no cleaning or disinfecting solutions will be used for this lens type.</li> <li>If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day between visits. One missed day of lens wear between visits is acceptable.</li> <li>Subjects will be instructed to wear study lenses to the next visit. It is not required that they have worn lenses for 6 hours on the day of the visit.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>Subjects will be instructed to bring their own spectacles or contact lenses to the</li> </ul> |

| Visit 2: Treatment 1 Follow-Up 1 | | |
|---|---|---|
| Step | Procedure | Details |
| | | next visit, if needed for exit distance |
| | | visual acuity measurement. |
| 2.29 | Schedule | The subject will be scheduled to return for |
| | Follow-up | their follow-up appointment in 7±1 days. |

VISIT 3

The subjects must present to Visit 3 wearing the study lenses.

| | Visit 3: Treatment 1 Follow-Up 2 | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 3.1. | Adverse Events and<br>Concomitant<br>Medications Review | Review any changes to the subject's medical history or concomitant medications from the previous study visit. Record any changes, and any adverse events. | |
| 3.2. | Wear time and<br>Comfortable Wear<br>time (Study Lenses) | Record the average wearing time and comfortable wearing time with the study lenses. | |
| 3.3. | Compliance | Confirm compliance with the prescribed wear schedule. | |
| 3.4. | Collect unworn<br>study lenses (if<br>applicable) | Any remaining unworn study lenses will be collected from the subject. | |
| 3.5. | PRO (CLUE and<br>MRD)<br>Questionnaires | The subject will respond to the Follow-Up PRO (CLUE and MRD) Questionnaires. | |
| 3.6. | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | |
| 3.7. | Subjective<br>Acceptance | Record whether the subject's distance and near vision with the lenses is acceptable. | |
| 3.8. | Entrance Distance<br>and Near Visual<br>Acuity | Record the distance and near Snellen visual acuity (OD, OS, OU) to the nearest letter with the study contact lenses in place. For near measurements use the ETDRS 2000 Series Chart 1 or 2. | |
| 3.9. | Binocular Distance<br>Over-refraction and<br>Distance Visual<br>Acuity | Perform a binocular over-refraction and record the OD and OS results and distance visual acuity. Note: No lens changes are allowed based on the over-refraction. | Appendix<br>G |
| 3.10. | Toric Fit Evaluation | Record: | |

| Visit 3: Treatment 1 Follow-Up 2 | | |
|---|---|---|
| Step | | |
| | | <ul> <li>The rotational position to the nearest degree</li> <li>Lens stability with blink</li> <li>Toric fit acceptable or unacceptable</li> </ul> |
| | | Toric lens fit will be unacceptable if lenses rotated more than 30 degrees, or lens stability is worse than 5 degrees movement with blink. If toric fit is unacceptable for either eye, the subject will be discontinued from the study. Remove and discard the lenses, then proceed to Final Evaluation. |
| 3.11. | Lens Fit Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). Lens fit will be unacceptable if any of the following is observed: • presence of limbal exposure (appearance of clear cornea) in any gaze • presence of edge lift • presence of excessive movement with blink in primary gaze • presence of insufficient movement in all three movement categories (primary gaze, upgaze, and push-up test). If lens fit is unacceptable for either eye, the subject will be discontinued from the study. Remove and discard the lenses, then proceed |
| 3.12. | Visual Performance<br>Distance (4 M)<br>Intermediate (64 cm)<br>Near (40 cm) | to Final Evaluation. Visual performance will be recorded OD, OS, and OU for the following: Distance, Bright Illuminance ETDRS Charts 4 M-HC#1, HC#2, HC#3 and LC#1, LC#2 and LC#3 Near, Bright Illuminance Reduced Guillon-Poling Charts High Contrast and Low Contrast Intermediate (64 cm) and Near (40 cm). |

| Visit 3: Treatment 1 Follow-Up 2 | | |
|---|---|---|
| Step | tep Procedure Details | |
| | | Distance, Dim Illuminance (with <u>Distance</u> goggles) ETDRS Charts 4 M-HC#4, HC#5, HC#6 Near, Dim Illuminance (with <u>Near</u> goggles) Reduced Guillon-Poling charts High Contrast Intermediate (64 cm) and Near (40 cm). Note: • The room illuminance must be between 7.3 and 7.9 EV (or 400 to 600 lux). • Distance, HC-1 Chart luminance Acceptable EV Range is 10.5-10.7 (or 180 to 210 cd/m²). • Guillon-Poling, Near Chart Luminance Acceptable EV Range is 10.8-11.1 (or 220 to 280 cd/m²). |
| | | luminance (Dim luminance will be |
| 2.12 | T D 1 | simulated by using the goggles). |
| 3.13. | Lens Removal | Have the subject remove the study lenses. Temporarily store the worn lenses until Biomicroscopy has been completed. If no adverse event or PQC was recorded, the worn lenses may be discarded. |
| 3.14. | Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings. If the clearance of the fluorescein needs to be expedited, preservative-free saline may be instilled. If the subject has a Grade 3 or worse slit lamp finding, it will be recorded as an Adverse Event and the subject will be monitored as per the guidelines given in section 13. |

#### FINAL EVALUATION

The final evaluation will ordinarily take place immediately following the last scheduled follow-up visit per the study protocol. It may also take place at any point the subject discontinues the study or is terminated from the study.

| | Final Evaluation | |
|---|---|---|
| Step | Procedure | Details |
| F.1 | Final Exam Form | Indicate if the subject completed the study successfully. If subject discontinued from the study, indicate the reason. |
| F.2 | Biomicroscopy (for<br>subjects that are<br>discontinued early) | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. If the clearance of the fluorescein needs to be expedited, preservative-free saline may be instilled. If the subject has a Grade 3 or worse slit lamp finding, it will be recorded as an Adverse Event and the subject will be monitored as per the guidelines given in section 13. |
| F.3 | Subjective<br>spherocylindrical<br>Refraction | An optimal, binocular balanced distance sphero-cylindrical refraction will be performed. Record the refraction and distance visual acuity (OD, OS, OU) to the nearest letter. |
| F.4 | Exit Distance Visual<br>Acuity | Record the distance Snellen visual acuity (OD, OS, OU) to the nearest letter, and the type of visual correction being worn (habitual lenses, distance spectacles or unaided). |

#### 7.3. Unscheduled Visits

If, during the investigation, a subject requires an unscheduled visit to the clinical site, the following information will be collected at a minimum:

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the adverse event must be completed and subject record completed as appropriate
- Date and time of the visit and all procedures completed at the unscheduled visit
- Review of adverse event and concomitant medications
- Documentation of any test article dispensed or collected from the subject, if applicable
- Slit lamp findings (using the Slit Lamp Classification Scale)

If the Investigator withdraws a subject from the study, the final study visit case report forms must be completed indicating the reason(s) why the subject was withdrawn. The subject record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that are ongoing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pre-

treatment status, stabilized, or been satisfactorily explained. If further treatment i.e., beyond licensure is required, the subject will be referred to the appropriate health care provider.

The following information will be collected during an unscheduled visit.

| Unscheduled Visit | | |
|---|---|---|
| Step | Procedure | Details |
| U.1 | Reason for | Indicate if the <u>only</u> reason for the visit is that |
| | unscheduled visit | the subject requires additional test articles. If |
| | | the reason is other than resupply of |
| | | previously dispensed lenses, specify the |
| | | reason for the visit. |
| U.2 | Chief Complaints (if | Record the subject's chief complaints for |
| | applicable) | reasons for the unscheduled visit. |
| U.3 | Adverse Events and | Review any changes to the subject's medical |
| | Concomitant | history or concomitant medications from the |
| | Medications Review | previous study visit. Record any changes, and |
| | (if applicable) | any adverse events. |
| U.4 | Entrance VA (if | Record the distance Snellen visual acuity |
| | applicable) | (OD, OS, OU) to the nearest letter, and the |
| | , | type of visual correction being worn (study |
| | | lenses, habitual lenses, distance spectacles or |
| | | unaided). |
| U.5 | Subjective Sphero- | Perform bare-eye subjective spherocylindrical |
| | cylindrical | refraction with a phoropter (adopt the |
| | Refraction (if | maximum plus to maximum visual acuity |
| | applicable) | (MPMVA) approach and use the duo-chrome |
| | | test for binocular balancing) and record the |
| | | best corrected <u>distance</u> visual acuity to the |
| | | nearest letter (OD, OS). |
| U.6 | Slit Lamp | FDA Slit Lamp Classification Scale will be |
| | Biomicroscopy (if | used to grade the findings. If the clearance of |
| | applicable) | the fluorescein needs to be expedited, |
| | | preservative-free saline may be instilled. |
| U.7 | Dispensing (if | If the subject requires additional lenses to |
| | applicable) | complete the wear period and is eligible to do |
| | | so, provide additional lenses per the |
| | | dispensing instructions given in the detailed |
| | | study procedures. |
| U.8 | Toric Fit | After lens settling, record: |
| | Evaluation (if | The rotational position to the nearest |
| | applicable) | degree |
| | | Lens stability with blink |
| | | · |
| | | Lens stability with eye versions |

| | Unscheduled Visit | |
|---|---|---|
| Step | Procedure | Details |
| | | Toric fit acceptable or unacceptable |
| | | Toric lens fit will be unacceptable if lenses |
| | | rotated more than 30 degrees, or lens |
| | | stability is worse than 5 degrees movement |
| | | with blink. If toric fit is unacceptable for |
| | | either eye, the subject will be discontinued |
| | | from the study. Remove and discard the |
| | | lenses, then proceed to Final Evaluation. |
| U.9 | Lens Fit Assessment (if applicable) | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). |
| | | Lens fit will be unacceptable if any of the |
| | | following is observed: |
| | | presence of limbal exposure (appearance |
| | | of clear cornea) in any gaze |
| | | presence of edge lift |
| | | presence of excessive movement with |
| | | <ul> <li>blink in primary gaze</li> <li>presence of insufficient movement in all</li> </ul> |
| | | three movement categories (primary gaze, |
| | | upgaze, and push-up test). |
| | | If lens fit is unacceptable for either eye, the |
| | | subject will be discontinued from the study. |
| | | Remove and discard the lenses, then proceed |
| U.10 | Exit Vigual Aquita | to Final Evaluation. |
| 0.10 | Exit Visual Acuity (if applicable) | Record the distance Snellen visual acuity (OD, OS, OU) to the nearest letter, and the |
| | (11 applicable) | type of visual correction being worn (study |
| | | lenses, habitual lenses, distance spectacles or |
| | | unaided). |

### 7.4. Laboratory Procedures

None

#### 8. SUBJECTS COMPLETION/WITHDRAWAL

#### 8.1. Completion Criteria

Subjects are considered to have completed the study if they:

- provided informed consent.
- are eligible.
- completed all visits

#### 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the study for any of the following reasons:

- Subject death during the study period.
- Subject withdrawal of consent.
- Subject not compliant to protocol
- Subject lost to follow-up.
- Subject no longer meets eligibility criteria (e.g., the subject becomes pregnant).
- Subject develops significant or serious adverse events causing discontinuation of study lens wear.
- Subjects who have experienced a Corneal Infiltrative Event (CIE).
- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment).
- Subject not compliant with study lens wear schedule.
- Subject not successfully dispensed due to lack of efficacy and safety including poor vision, poor comfort or unacceptable fit.

For discontinued subjects, the Investigator will:

- Complete the current visit (scheduled or unscheduled).
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study.
- Record the spherocylindrical refraction with best corrected distance visual acuity.
- Collect used test article(s) (worn or brought to the visit) from the subject and discard them, unless otherwise stated in Section 7.2.
- Collect all unused test article(s) from the subject.
- Make arrangements for subject care, if needed, due to their study participation

An additional subject may be enrolled if a subject discontinues from the study prematurely.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

#### 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Disallowed medications and therapies are medications or therapies that contraindicate contact lens wear. See the Exclusion criteria for specific details.

#### 9.1. Systemic Medications

Certain systemic medications are known to have a higher likelihood to interfere with contact lens wear, chiefly by disrupting the tear film. A summary of disallowed medications is shown in Table 4. Subjects with a history of taking these medications will be allowed to enroll only if:

 The medications have been taken on a continual or routine basis for at least 6 months and the subject has demonstrated successful contact lens wear during this time.

Or

 The subject previously used these medications on a temporary basis and has ceased that medication at least 1 week prior to signing the informed consent.

Table 4: Disallowed systemic medications

| Class of Drug | Common Indication(s) | Common Examples |
|---|---|---|
| Anticholinergics | Irritable bowel syndrome, Parkinson's disease, peptic ulcer, cystitis, nasal congestion, cold symptoms, overactive bladder, COPD | Bentyl, Spiriva, Atrovent,<br>Hyosyne, Levsin, Symax<br>Fastab, Symax SL, Homax SL,<br>Cogentin, Transderm Scop, etc. |
| Oral Phenothiazines | Antipsychotic disorders (schizophrenia, mania) | Compazine, Mellaril,<br>Thorazine, Phenergan, etc. |
| Oral/Inhaled<br>Corticosteroids | Arthritis, colitis, asthma,<br>bronchitis, allergic or<br>inflammatory conditions | Cortisone, Prednisone,<br>Hydrocortisone, Medrol,<br>Kenalog, Flonase etc. |
| Oral Retinoids | Seborrhea, acne | Isotretinoin, Acitretin,<br>Alitretinoin, etc. |
| Oral Tetracycline | Urinary Tract Infection, acne,<br>chlamydia, gonorrhea | Sumyein, Achromyein V, etc. |

#### 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Protocol deviations must be reported to the sponsor within 24 hours after discovery of the protocol deviation. The Investigator will report deviations per IRB/IEC requirements. All deviations will be tracked, and corrective actions implemented as appropriate.

If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigator must notify and provide the rationale to the Sponsor and, as required, the IEC/IRB.

If the deviation potentially impacts the safety of patient or changes the technical integrity of the study, then it must be reported to IEC/IRB. This is a "Major Deviation". Deviations that contradict the information contained in the Informed Consent/Assent forms will be considered Major Deviations.

Minor deviations have no substantive effect on patient safety or technical integrity of the study. They are often logistical in nature.

Protocol waivers are prohibited.

Table 5 lists examples of deviations that will constitute major and minor protocol deviations for this study.

Table 5: Examples of major and minor protocol deviations

| Deviation category | Major deviation | Minor deviation |
|---|---|---|
| Out-of-window visit | Visit attended 3 or more days<br>out of visit window defined<br>in study procedures | Visit attended 2 or fewer days out of visit window defined in study procedures |
| Insufficient wear of study lenses | Subject does not wear study lenses for at least 6 hours per day for 3 or more days between scheduled visits. | Subject does not wear study lenses for at least 6 hours per day for 2 days between scheduled visits. |
| Unanswered PRO questions | For questionnaires where data is related to a primary or secondary endpoint, more than 2 PRO questions are unanswered (i.e., left blank). | For questionnaires where data is related to a primary or secondary endpoint, 2 or fewer PRO questions are unanswered (i.e., left blank). For questionnaires where data is not related to a primary or secondary endpoint, any PRO questions are unanswered (i.e., left blank). |

#### 11. STUDY TERMINATION

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further dispensing of test article. In the event of a USADE or SAE, the Sponsor will discuss this with the Investigator before any further subjects are enrolled.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if information indicates the study's results are compromised.

JJVC reserves the right to terminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to specific clinical observations, if in their opinion, after a discussion with JJVC, it is determined that it would be unwise to continue at the clinical site.

JJVC (and the IEC/IRB, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

#### 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

- Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)."
- Clinical test articles that are stored improperly or damaged after receipt at the investigational site.
- Lens replacements that occur due to drops/fall-outs.
- Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency (i.e. tears, rips, etc.), only in situations where there is no deficiency alleged by the subject.

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use

is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness).
- Who received the complaint.
- Study number.
- Clinical site information (contact name, site ID, telephone number).
- Lot number(s).
- Unique Subject Identifier(s).
- Indication of who first observed complaint (site personnel or subject).
- OD/OS indication, along with whether the lens was inserted.
- Any related AE number if applicable.
- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.).
- Eye Care Provider objective (slit lamp) findings if applicable.
- Confirmation of product availability for return (and tracking information, if available), or rationale if product is not available for return

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow Section 13 of this protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also apply and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

**Adverse Event (AE)** – An AE is "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device."

**Note**: This definition includes events related to the investigational medical device or the comparator, and to the procedures involved. For users or other persons, this definition is restricted to events related to investigational medical devices.

An AE includes any condition (including a pre-existing condition) that:

- 1. Was not present prior to the study, but appeared or reappeared following initiation of the study.
- 2. Was present prior to the study but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states.

**Note**: Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event.

Serious Adverse Event (SAE) – An SAE is any adverse event that led to any of the following:

- Death
- Serious deterioration in the health of the subject that resulted in any of the following:
  - Life-threatening illness or injury
  - o Permanent or persistent impairment of a body structure or a body function
  - o Hospitalization or prolongation of patient hospitalization
  - Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.
  - o Chronic disease
- Foetal distress, foetal death or a congenital physical or mental impairment of birth defect.

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization
- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect
- Limbal cell Damage leading to Conjunctivalization

**Significant Adverse Events** – are defined as events that are symptomatic and warrant discontinuation (temporary or permanent) of the contact lens wear

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)

- Any Temporary Loss of > 2 Lines of BSCVA
- Other grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation > 2 weeks

**Non-Significant Adverse Events** – are defined as those events that are usually asymptomatic and usually do not warrant discontinuation of contact lens wear but may cause a reduction in wear time. However, the Investigator may choose to prescribe treatment as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis
- Localized Allergic Reactions
- Hordeolum
- Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation < 2 weeks

**Adverse Device Effect (ADE)** – An ADE is an "adverse event related to the use of an investigational medical device."

**Note 1**: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.

**Note 2**: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device.

**Note 3:** This includes 'comparator' if the comparator is a medical device. <sup>1</sup>

**Serious Adverse Device Effect (SADE) -** Any adverse device effect that has resulted in any of the consequences characteristic of a serious adverse event.

Unanticipated Serious Adverse Device Effect (USADE): serious adverse device effect (SADE) which by its nature, incidence, severity or outcome has not been identified in the current risk assessment.

**Note 1:** USADE is synonymous with UADE below from the United States (US) Code of Federal Regulations (CFR).

**Note 2:** Anticipated serious adverse device effect (ASADE) is an effect which by its nature, incidence, severity or outcome has been identified in the risk assessment.

Unanticipated Adverse Device Effect (UADE) – A UADE is any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects.

**Note 1**: UADE is synonymous with USADE above from ISO 14155.

#### 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in section 13.1).
- Causality or Relatedness i.e. the relationship between the test article, study treatment or study procedures and the adverse event (not related, unlikely related, possibly related, or related see definition in Section 13.2.1).
- Adverse Event Severity Adverse event severity is used to assess the degree of intensity of the adverse event (mild, moderate, or severe see definition in Section 13.2.2).
- Outcome not recovered or not resolved, recovering or resolving, recovered or resolved with sequelae, recovered or resolved, death related to adverse event, or unknown.
- Actions Taken none, temporarily discontinued, permanently discontinued, or other.

#### 13.2.1. Causality Assessment

Causality Assessment – A determination of the relationship between an adverse event and the test article, study treatment, or the study procedures. The test article, study treatment, or study procedures relationship for each adverse event should be determined by the investigator using these explanations:

- Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures.
- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely.
- Possibly Related An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g. concomitant treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded.
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g. concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge and re-challenge.

#### 13.2.2. Severity Assessment

**Severity Assessment** – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

- Mild Event is noticeable to the subject but is easily tolerated and does not interfere with the subject's daily activities.
- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities.
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the subject's daily activities.

#### 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begin when the subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs and complete the Adverse Event eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

- Adverse event (diagnosis not symptom).
- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.).
- Date the clinical site was notified.
- Date and time of onset.
- Date and time of resolution.
- Adverse event classification, severity, and relationship to test articles, as applicable.
- Treatment regimen instituted (where appropriate), including concomitant medications prescribed, in accordance with applicable licensing requirements.
- Any referral to another health care provider if needed.
- Outcome, ocular damage (if any).
- Likely etiology.

• Best corrected visual acuity at the discovery of the event and upon conclusion of the event, if the AE is related to the visual system.

Upon discovery of an AE that is deemed 'possibly related' or 'related' to the test article or study procedures (whether related to the visual system or not), an AE review form must be completed. Additional dated and initialed entries should be made at follow-up evaluations. Separate forms must be completed for each eye if the AE is bilateral.

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the Test Article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the subject will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date, should be followed to resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator. Non-ocular adverse events that are not related to the test article, study treatment, or study procedures may be recorded as "ongoing" without further follow-up.

#### 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by EDC System, e-mail, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition, a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (Section 13.4.2). The report will comment whether the adverse event was considered to be related to the test article, study treatment or study procedures.

#### 13.4.1. Reporting Adverse Events to Sponsor

#### **Serious/Significant Adverse Events**

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by EDC system, e-mail or telephone, but no later

than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

In the event of a serious/significant adverse event, the Investigator must:

- Notify the Sponsor immediately.
- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject.
- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article.
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations.

#### **Unanticipated (Serious) Adverse Device Effect (UADE)**

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

#### **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

#### 13.4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according to the written guidelines, including reporting timelines.

#### 13.5. Event of Special Interest

None

#### 13.6. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant subjects and their fetuses

will not be monitored for study related purposes. Pregnant subjects are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

#### 14. STATISTICAL METHODS

#### 14.1. General Considerations

Statistical Analysis will be undertaken by the sponsor or under the authority of the sponsor. A general description of the statistical methods to be implemented in this clinical trial is outlined below. More details will be included in the stand-alone Statistical Analysis Plan (SAP). The SAP will be developed and finalized prior to database lock.

Data manipulation, statistical summaries and statistical analyses will be performed using the Statistical Analysis System (SAS) software Version 9.4 or higher (SAS Institute, Cary, NC)<sup>11</sup>.

Descriptive statistics will be reported for all key variables as appropriate. Continuous data will be summarized descriptively by sample size (n), mean, standard deviation (SD), median, minimum (Min) and maximum (Max). Categorical data will be summarized descriptively by frequency count (n) and percentage (%) of subjects or eyes within each category level. Summary tables will be presented by event (Baseline, Fitting, 1-Week follow-up, 2-Week follow-up, Unscheduled and Final Evaluations) and study lens type as applicable, for the analysis set of interest. The denominator for all percentages will be the number of subjects (or eyes, as applicable) with available data in the lens group under consideration. Unscheduled visits and tele-visits will be summarized separately and will be excluded from the co-primary and secondary efficacy analyses.

#### 14.2. Sample Size Justification

The total sample size of 140 subjects who complete the study (Visit 3) was calculated to provide adequate power in detecting statistical superiority of the Test lens relative to prespecified thresholds for binocular distance, intermediate and near logMAR VA, CLUE vision Scores, Absolute toric rotation, rotational stability, rate of unacceptable lens fitting and rate of grade 3 or higher SLFs. All co-primary effectiveness and safety hypotheses are required to achieve statistical significance for the study objective to be satisfied, therefore no adjustment for multiple primary hypotheses is necessary. Each co-primary hypothesis will be tested using a 1-sided Type I error rate of 0.025.

Thresholds for hypotheses associated with CLUE vision, comfort and, handling scores are from a meta-analysis of 14 JJVCI clinical trials of toric and multifocal toric contact lenses used by habitual contact lens wearers aged 40 to 70 years<sup>12</sup>. In this analysis, baseline CLUE scores (for subjects' habitual contact lenses) from 14 clinical studies were analyzed to establish thresholds reflecting the "real-world" performance of contact lenses wearers in this population

with respect to CLUE vision, comfort, and handling scores. Thresholds for all other endpoints were based on clinically relevant margins.

Additionally, this study was also powered to test superiority for secondary endpoints with respect to CLUE vision, comfort and, handling scores and lens fit success using a 1-sided Type I error rate of 0.025. Secondary endpoints will be tested using a fixed sequence approach. Further details on the preservation of the study overall Type I error rate are in Section 14.4.

The sample size of 140 to complete yields at least 81% overall power to detect statistical superiority for all co-primary endpoints. This sample size provides a statistical power of at least 99% for each co-primary and secondary endpoint. To account for subject drop-out approximately 155 subjects will be enrolled to ensure at least 140 subjects complete the study.

Table 6: Sample Size Estimates by Study Endpoint

| Endpoint<br>Domain | Endpoint | Statistical Test Type<br>(Statistically<br>Significantly) | Sample<br>Size | Power (%) |
|---|---|---|---|---|
| Primary<br>Efficacy | Distance (4m) Binocular Visual<br>Acuity (logMAR) | Superiority: mean VA< 0.00 | 9 | 99.1 |
| | Intermediate (64cm) Binocular<br>Visual Acuity (logMAR) | Superiority: mean VA< 0.17 | 6 | 99.5 |
| | Near (40cm) Binocular Visual<br>Acuity (logMAR) | Superiority: mean VA< 0.17 | 29 | 99.1 |
| | CLUE Vision Scores - Myopes | Superiority: mean score> 41 | 29 | 99.2 |
| | CLUE Vision Scores - Hyperopes | Superiority: mean score> 36 | 23 | 99.0 |
| | Absolute Toric Rotation ≤ 10° | Superiority: percentage>80% | 140 | >99 |
| | Lens Stability with Blinks ≤ 5° | Superiority: percentage>80% | 140 | 96.8 |
| Primary<br>Safety | Grade 3 or Higher SLFs (%) | Superiority: percentage< 5% | 140 | 89.3 |
| | Unacceptable Lens Fitting (%) | Superiority: percentage<20% | 140 | >99 |
| Secondary | CLUE Handling Scores: Hyperopes | Superiority: mean score> 46 | 15 | 99.2 |
| Efficacy | CLUE Comfort Scores - Hyperopes | Superiority: mean score> 38 | 23 | 99.2 |
| | CLUE Vision Scores - Hyperopes | Superiority: mean score> 41 | 42 | 99.1 |
| | CLUE Handling Scores - Myopes | Superiority: mean score> 55 | 26 | 99.1 |
| | CLUE Comfort Scores - Myopes | Superiority: mean score> 51 | 46 | 99.1 |
| | CLUE Vision Scores - Myopes | Superiority: mean score> 46 | 55 | 99.0 |
| | Lens Fit Success Rate (%) | Superiority: percentage>90% | 140 | 99.8 |

This will be the first dispensing study since the lens design was changed hence, historical clinical data on the previous lens design has been used for the sample size calculations for any of the study endpoints except for toric rotation and lens stability with blinks. The changes made to the lens design improved the rotational performance of the contact lens and were not considered to impact the visual acuity or the subjective performance of the lens. Sample size estimates for toric rotation and lens stability with blinks were calculated using the results from

study while the sample size estimates for all other efficacy endpoints utilized data from study Historical data for each endpoint is summarized in Table 7 below.

Table 7: Historical Data by Endpoint

| | | Value: Mean (SD) or |
|---|---|---|
| Endpoint Type | Endpoint | Percentage of Eyes |
| | Distance Binocular logMAR VA | -0.13 (0.078) |
| | Intermediate Binocular logMAR VA | -0.05 (0.092) |
| | Near Binocular logMAR VA | 0.07 (0.120) |
| *Primary Efficacy Endpoints | Vision Scores – Hyperopes | 54.32 (19.506) |
| | Vision Scores – Myopes | 57.97 (20.282) |
| | Absolute Toric Rotation ≤ 10° | 90.20% |
| | Lens Stability with Blinks ≤ 5° | 100% |
| *Secondary Efficacy | Handling Scores - Hyperopes | 67.52 (17.665) |
| Endpoints | Handling Scores - Myopes | 71.48 (18.578) |
| | Comfort Scores - Hyperopes | 57.95 (20.864) |
| | Comfort Scores - Myopes | 64.97 (21.479) |
| | Lens Fit Success | 100% |
| **Primary Safety Endpoints | Unacceptable Lens Fitting | 0.0% |
| | Grade 3+ SLFs (Ocular Adverse Events) | 0.0% |

SD: Standard Deviation

#### Co-Primary Efficacy Endpoint Sample Size Calculations:

#### Distance, Intermediate and, Near logMAR Visual Acuity

Sample size calculations for distance, intermediate and near visual acuity were carried out separately using one-sided, one-sample mean t-test, with a one-sided Type I error rate of 0.025 for each hypothesis using the *One-Sample T-Tests for Superiority by a Margin* procedure in Power Analysis & Sample Size (PASS2021) software Version 21.0.6 (NCSS LLC, Kaysville UT)<sup>13</sup>. To preserve the overall study power, each endpoint was powered to approximately 99%. The assumptions for averages and standard deviations were made based on historical values from previous studies (Table 7).

#### CLUE Vision Scores (Hyperopes and Myopes)

Sample size calculations for CLUE Vision scores were carried out separately for each sphere stratum (hyperopes and Myopes) using one-sided, one-sample mean t-test, with a one-sided Type I error rate of 0.025 for each hypothesis using the *One-Sample T-Tests for Superiority by a Margin* procedure in Power Analysis & Sample Size (PASS2021) software Version 21.0.6 (NCSS LLC, Kaysville UT)<sup>13</sup>. To preserve the overall study power, each endpoint was powered to approximately 99%. The assumptions for averages and standard deviations were made based on historical values from previous studies (Table 7).

<sup>\*</sup>Summaries for primary efficacy and secondary endpoints were provided for the per-protocol population at the 1-week follow-up evaluation.

<sup>\*\*</sup>Summaries for the primary safety endpoints were provided for the safety population; all available data was included

#### Toric Rotation and Lens Stability

The reference rate for absolute toric lens rotation  $\leq 10^{\circ}$  was based on the historical results of 90.2%. The reference rate for lens stability  $\leq 5^{\circ}$  was based on the worst-case scenario of 99%, given the historical results show 100%. Toric lens orientation and rotational stability, respectively, are defined as a binary response:

$$Toric \ Lens \ Orientation: Y \\ = \begin{cases} 1 & \text{if a subject eye has absolute toric lens rotation} \leq 10^{\circ} \\ 0 & \text{Otherwise} \end{cases},$$
 
$$Rotational \ stability: Z = \begin{cases} 1 & \text{if a subject eye has lens stability with blinks} \leq 5^{\circ}, \\ 0 & \text{Otherwise} \end{cases}$$

Historical data of the Test lens indicates there is a high rate ( $\geq 90\%$ ) for both toric lens rotation  $\leq 10^\circ$  and rotational lens stability. Assuming a correlation of 0.70 between left and right eyes, a total of 5000 replicating trials were simulated with reference rate of 90.2% for the percentage of eyes with small ( $\leq 10^\circ$ ) absolute toric lens rotation (or 99% of eyes with rotational stability). Given the high event rate of the binary outcome, Y=1, each replicated sample was analyzed using a Bayesian beta-binomial model with correlated binary data (Diniz et al; 2010)<sup>14</sup>. A non-informative prior distribution, beta (0.5, 0.5) was used to model  $P_T$  (proportion of eyes with absolute toric lens rotation  $\leq 10^\circ$  [or lens stability  $\leq 5^\circ$ ] for the Test lens). For each simulated trial, the 95% central posterior credible interval (CrI) constructed for the percentage of eyes with absolute toric lens rotation  $\leq 10^\circ$  [or lens stability  $\leq 5^\circ$ ] for the Test lens was calculated. The null and alternative hypothesis for determining statistical significance in both endpoints were  $P_T \leq 80\%$  and  $P_T > 80\%$ , respectively. With the proposed sample size, each endpoint (percentage of eyes with absolute toric lens rotation  $\leq 10^\circ$  and lens stability  $\leq 5^\circ$ ) has at least 96% power, i.e., 96% of the estimated 95% CrIs had the lower bound above 80%.

#### **Co-Primary Safety Endpoint Sample Size Calculations:**

#### Grade 3 or Higher Slit Lamp Findings (SLF) and Unacceptable Lens Fitting

Grade 3 or Higher SLFs related to study lens wear was converted to a binary response as Y=1, if a subject eye has a clinically significant SLF, and Y=0 otherwise, for analysis purposes. Historical data show none or an extremely low rate (<1%) for clinically significant SLFs (Grade 3 or higher) for the test lens. Assuming a correlation of 0.70 between left and right eyes, a total of 5000 replicating trials were simulated with a reference rate of 1% (worse-case scenario). Given the rare event binary outcome of slit lamp findings, each replicated sample was analyzed using a Bayesian beta-binomial model with correlated binary data (Diniz et al;  $2010)^{14}$ . A non-informative prior distribution, beta (0.5, 0.5) was used to model  $P_T$  (proportion of eyes with Grade 3 or higher SLF for the Test lens). For each simulated trial, the 95% central posterior credible interval constructed for the percentage of eyes with grade 3 or higher SLFs for the Test lens was calculated. The null and alternative hypothesis for statistical significance

were  $P_T \ge 5\%$  and  $P_T < 5\%$ , respectively. With the proposed sample size, at least 99% of the estimated 95% credible intervals had the upper bound below 5%.

As indicated in Table 6, co-primary safety endpoints were powered to at least  $\sim$ 89% individually, yielding a combined power of  $\sim$ 88%. With respect to co-primary efficacy, each hypothesis, was powered to  $\sim$ 99%, which provided a combined power of  $\sim$ 92%. Therefore, the overall combined study power for co-primary safety and co-primary efficacy hypotheses is  $\sim$ 81%.

#### **Secondary Efficacy Endpoint Sample Size Calculations:**

#### CLUE Vision, Comfort and, Handling (Hyperopes and Myopes)

Sample size calculations for the secondary endpoints of CLUE vision, comfort, and handling scores were carried out separately for each sphere stratum (hyperopes and Myopes) for all three CLUE domains using one-sided, one-sample mean t-test, with a one-sided Type I error rate of 0.025 for each hypothesis using the *One-Sample T-Tests for Superiority by a Margin* procedure in Power Analysis & Sample Size (PASS2021) software Version 21.0.6 (NCSS LLC, Kaysville UT)<sup>13</sup>. The assumptions for averages and standard deviations were made based on historical values from previous studies (Table 7).

#### Lens Fit Success

The reference rate for lens fit success was based on the worst-case scenario of 99%, given the historical results show 100% (Table 6). Lens fit is a binary response and is defined as follows:

Lens Fit Success: 
$$Y = \begin{cases} 1 & \text{if a subjects'} vision is optimized in 2 pairs or less} \\ 0 & \text{Otherwise} \end{cases}$$

Historical data of the Test lens indicates there is an extremely high rate (100%) for lens fit success. Assuming a correlation of 0.70 between left and right eyes, a total of 5000 replicating trials were simulated with reference rate of 99% for the percentage of eyes optimized in 4 lenses (2 pairs) or less. Given the high event rate of the binary outcome, Y=1, each replicated sample was analyzed using a Bayesian beta-binomial model with correlated binary data (Diniz et al; 2010)<sup>14</sup>. A non-informative prior distribution, beta(1, 1) was used to model  $P_T$  (proportion of eyes with optimized in 4 lenses or less). For each simulated trial, the 95% central posterior credible interval (CrI) constructed for the percentage of eyes optimized in 4 lenses or less was calculated. The null and alternative hypothesis for determining statistical significance were  $P_T \le 90\%$  and  $P_T > 90\%$ , respectively. With the proposed sample size, the percentage of eyes optimized in 4 lenses or less has at least 99% power, i.e., 99% of the estimated 95% CrIs had the lower bound above 90%.

#### 14.3. Analysis Populations

#### **Safety Population:**

All subjects who were administered any test article.

#### **Per-Protocol Population:**

All subjects who have successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock (Per-Protocol Population). Justification of excluding subjects with protocol deviations will be documented in a memo to file.

#### **Intention-to-Treat (ITT) Population:**

Intention-to-treat population will include all assigned subjects.

#### 14.4. Level of Statistical Significance

The Type I error rate of the trial will be controlled at 1-sided 0.025 level. Each co-primary safety and efficacy hypothesis will be tested using a 1-sided Type I error of 0.025. All co-primary hypotheses must be met to satisfy the study objectives and to test any secondary hypotheses.

Based on a gate keeping approach between the primary and secondary families of hypotheses, all primary endpoints must show statistical significance at one-sided 0.025 level in order to pass the full alpha level to test the secondary endpoints hypotheses.

A fixed sequence testing procedure will be utilized to test the secondary hypotheses to control the Type I error rate also in the secondary family of hypotheses. Each secondary hypotheses will be tested using a 1-sided 0.025 level following the order prespecified in section 2.3.3. Based on the fixed sequence principle, each secondary endpoint must be found statistically significant at a one-sided 0.025 level in order to proceed to the next step. If not, the testing procedure of the secondary endpoints will stop.

#### 14.5. Primary Analysis

The co-primary efficacy analyses will be conducted on the ITT population, while co-primary safety analyses will be conducted on the safety population. All efficacy and safety analyses will be based on observed case data with no imputation of missing values.

#### 14.5.1. Co-Primary Efficacy Analyses

#### Binocular HLHC Distance, Intermediate and, Near LogMAR Visual Acuity

Binocular, high luminance, high contrast visual acuity on logMAR scale after approximately 2-Weeks in the optimized lenses will be analyzed using a linear mixed model. Distance (distance/intermediate/near), sphere strata (hyperope and myope) and the interaction between distance by sphere strata will be included as fixed effects. Other baseline characteristics, such as age, gender and add power may be included as covariates when appropriate. Site will be

included as random effect (G-side). The covariance between residual errors from the same subject across distance will be modeled using an unstructured (UN) covariance structure. Mean estimates will be conducted using two-sided confidence intervals (CI) constructed for the least square mean. One-sided p-values will also be calculated.

The null and alternative hypothesis for binocular distance HLHC visual performance to test for superiority of the investigational lens relative to the pre-defined threshold of 0.00 logMAR is as follows:

$$H_o$$
:  $\mu_{Test} \ge 0.00 \log MAR$   
 $H_A$ :  $\mu_{Test} < 0.00 \log MAR$ 

Where  $\mu_{Test}$  represents the population mean for the investigational lens after 2-weeks lens wear with respect to distance binocular HLHC VA. The investigational lens will be declared statistically significantly lower than 0.00 logMAR if the one-sided p-values is below 0.025.

The null and alternative hypothesis for binocular intermediate HLHC visual performance to test for superiority of the investigational lens relative to the pre-defined threshold of 0.17 logMAR is as follows:

$$H_o$$
:  $\mu_{Test} \ge 0.17 \log MAR$   
 $H_A$ :  $\mu_{Test} < 0.17 \log MAR$ 

Where  $\mu_{Test}$  represents the population mean for the investigational lens after 2-Weeks lens wear with respect to intermediate binocular HLHC VA. The investigational lens will be declared statistically significantly lower than 0.17 logMAR if the one-sided p-values is below 0.025.

The null and alternative hypothesis for binocular near HLHC visual performance to test for superiority of the investigational lens relative to the pre-defined threshold of 0.17 logMAR is as follows:

$$H_o$$
:  $\mu_{Test} \ge 0.17 \log MAR$   
 $H_A$ :  $\mu_{Test} < 0.17 \log MAR$ 

Where  $\mu_{Test}$  represents the population mean for the investigational lens after 2-weeks lens wear with respect to near binocular HLHC VA. The investigational lens will be declared statistically significantly lower than 0.17 logMAR if the one-sided p-values is below 0.025.

#### **CLUE Vision Scores**

CLUE Vision Scores after approximately 2-Weeks in the optimized lenses will be analyzed using a linear mixed model adjusting for baseline scores as a covariate. Strata (hyperope and myope) will be included as the only fixed effect. Other baseline characteristics known of importance such as age, gender and Additional (ADD) power may be included as covariates when appropriate. Site will be included as random effect (G-side). The Kenward and Roger method will be used for the calculation of the denominator of degrees of freedom<sup>15</sup>. Mean estimates will be conducted using two-sided confidence intervals (CI) constructed for the least square mean. One-sided p-values will also be calculated.

The null and alternative hypothesis to test for superiority of the myopic subjects relative to the pre-defined threshold of 41 for the investigational lens is as follows:

$$H_o$$
:  $\mu_{Myopes} \le 41$   
 $H_A$ :  $\mu_{Myopes} > 41$ 

Where  $\mu_{Myopes}$  represents the population mean for the investigational lens after 2-Weeks lens wear with respect to CLUE Visions scores for myopic subjects. The investigational lens will be declared statistically significantly greater than 41 if the one-sided p-values is below 0.025.

The null and alternative hypothesis to test for superiority of the hyperopic subjects relative to the pre-defined threshold of 36 for the investigational lens is as follows:

$$H_o$$
:  $\mu_{Hyperopes} \le 36$   
 $H_A$ :  $\mu_{Hyperopes} > 36$ 

Where  $\mu_{Hyperopes}$  represents the population mean for the investigational lens after 2-weeks lens wear with respect to CLUE Visions scores for hyperopic subjects. The investigational lens will be declared statistically significantly greater than 36 if the one-sided p-values is below 0.025.

#### Toric Lens Orientation and Rotational Stability at least 15-minutes Following Settling

Absolute toric lens orientation (degrees) will be dichotomized as Y = 1 if absolute toric lens rotation (degrees)  $\leq 10^{\circ}$ ) and Y = 0 otherwise. Rotational stability will be quantified by lens stability with blinks (degrees). Lens stability will be dichotomized as X = 1 if the lens stability with blinks (degrees)  $\leq 5^{\circ}$  and X = 0 otherwise.

Absolute toric lens orientation and rotational stability will be analyzed separately using a Bayesian beta-binomial model with correlated binary data<sup>14</sup>.

The Model:

Let Y (the percentage of eyes with grade 3 or higher SLFs) be the sum of equicorrelated binary responses ( $Y_1$  and  $Y_2$  denotes left and right eyes, respectively) with probability of success p and correlation coefficient  $\rho$ .

The probability distribution of  $Y = Y_1 + Y_2$  is obtained by the mixture of two variables. One of them follow a binomial distribution Bin(2, p) with probability of success p and mixing probability  $(1 - \rho)$ , and the other follows a modified Bernoulli distribution MBern(p), taking values 0 and 2, with probability of success p and mixing probability  $\rho$ :

$$P(Y = y | p, \rho) = (1 - \rho) Bin(2, p)I_{A1} + \rho MBern(p)I_{A2}$$

where  $I_{A1} = \{0, 1, 2\}$ ,  $I_{A2} = \{0, 2\}$  and p is the probability of success (i.e. proportion of eyes with Grade 3 or Higher SLFs).

To overcome the complexity of the mixture likelihood, a latent variable  $Z_i$ , i = 1, 2 is introduced in the model to indicate in which component of the correlated binary model the observation  $y_i$ , i = 1, 2 belongs to, that is,

$$Z_i = \begin{cases} 1 & \text{if the observation belong to } MBern(p) \\ 0 & \text{if the observation belong to } Bin(2, p) \end{cases}$$

The joint distribution of the augmented data  $(Y_i, Z_i)$ , i = 1, 2, is given by

$$P(Y = y_i, Z = z_i | p, \rho)$$

$$= \rho^{z_i} p^{\frac{y_i z_i}{2}} (1 - p)^{(2 - y_i)\frac{z_i}{2}} (1 - \rho)^{1 - z_i} {2 \choose y_i} p^{y_i (1 - z_i)} (1 - p)^{(2 - y_i)(1 - z_i)}$$

The probability p links to the regression variables through a logit transformation as follow:  $logit(p) = \beta_o + \beta_1 lens$ 

It is assumed that  $\beta_o$ ,  $\beta_1$  and  $\rho$  to be independent with a non-informative prior N(0, 1000) for  $\beta_o$  and  $\beta_1$ , and beta(0.5, 0.5) for  $\rho$ . The Metropolis sampler algorithm as implemented in the SAS/STAT MCMC procedure<sup>11</sup> will be used to estimate the posterior distributions of the parameters ( $\beta_o$ ,  $\beta_1$ ,  $\rho$ ). Inferences will be made based on a posterior credible interval for the relevant parameters.

The null and alternative hypotheses for evaluating superiority of the Test lens relative to 0.80 for are as follows:

$$H_o: p_T \le 80\%$$
  
 $H_1: p_T > 80\%$
where  $p_T$  is the percentage of eyes with absolute toric rotation  $\leq 10^\circ$  (or lens stability  $\leq 5^\circ$ ) for the investigational lens. Based on Bayesian posterior probability distribution of the proportion  $p_T$ , superiority is interpreted as 95% probability of the investigational lens being statistically higher than the threshold of 80% (i.e.,  $p_T > 80\%$ ). If the lower bound of the 95% central posterior credible interval is above 80%, it will be concluded that there is 95% probability that the investigational lens is statistically significantly higher than 80% based on observed sample.

# 14.5.2. Co-Primary Safety Analyses

The primary safety analyses will be conducted on the safety population.

# Grade 3 or Higher SLFs and Unacceptable Lens Fitting

Grade 3 of Higher SLFs (or Unacceptable lens fitting) will be analyzed using a Bayesian betabinomial model with correlated binary data<sup>14</sup>.

### The Model:

Let Y (the percentage of eyes with grade 3 or higher SLFs [or unacceptable lens fitting]) be the sum of equicorrelated binary responses ( $Y_1$  and  $Y_2$  denotes left and right eyes, respectively) with probability of success p and correlation coefficient p.

The probability distribution of  $Y = Y_1 + Y_2$  is obtained by the mixture of two variables. One of them follow a binomial distribution Bin(2, p) with probability of success p and mixing probability  $(1 - \rho)$ , and the other follows a modified Bernoulli distribution MBern(p), taking values 0 and 2, with probability of success p and mixing probability  $\rho$ :

$$P(Y = y | p, \rho) = (1 - \rho) Bin(2, p)I_{A1} + \rho MBern(p)I_{A2}$$

where  $I_{A1} = \{0,1,2\}$ ,  $I_{A2} = \{0,2\}$  and p is the probability of success (i.e. proportion of eyes with Grade 3 or Higher SLFs).

To overcome the complexity of the mixture likelihood, a latent variable  $Z_i$ , i = 1, 2 is introduced in the model to indicate in which component of the correlated binary model the observation  $y_i$ , i = 1, 2 belongs to, that is,

$$Z_i = \begin{cases} 1 & \text{if the observation belong to } MBern(p) \\ 0 & \text{if the observation belong to } Bin(2, p) \end{cases}$$

The joint distribution of the augmented data  $(Y_i, Z_i)$ , i = 1, 2, is given by

$$\begin{split} P(Y = y_i, Z = z_i | \, p, \rho) \\ &= \, \rho^{z_i} \, p^{\frac{y_i z_i}{2}} \, (1 - p)^{(2 - y_i) \frac{z_i}{2}} \, (1 - \rho)^{1 - z_i} \, \binom{2}{v_i} \, p^{y_i \, (1 - z_i)} \, (1 - p)^{(2 - y_i)(1 - z_i)} \end{split}$$

The probability p links to the regression variables through a logit transformation as follow:  $logit(p) = \beta_0 + \beta_1 lens$ 

It is assumed that  $\beta_o$ ,  $\beta_1$  and  $\rho$  to be independent with a non-informative prior N(0, 1000) for  $\beta_o$  and  $\beta_1$ , and beta(0.5, 0.5) for  $\rho$ . The Metropolis sampler algorithm as implemented in the SAS/STAT MCMC procedure<sup>11</sup> will be used to estimate the posterior distributions of the parameters ( $\beta_o$ ,  $\beta_1$ ,  $\rho$ ). Inferences will be made based on a posterior credible interval for the relevant parameters.

Bayesian Estimation and Statistical Evaluation of Hypothesis:

The null and alternative hypotheses for Grade 3 or higher SLFs of the investigational lens compared to the threshold of 5% are as follows:

$$H_o: p_T \ge 5\%$$
  
 $H_1: p_T < 5\%$ 

where  $p_T$  is the probability of a grade 3 or higher SLF across all study visits for test lens. Based on Bayesian posterior probability distribution of the proportion  $p_T$ , superiority is interpreted as 95% probability of test being statistically lower than the threshold of 5% (i.e.,  $p_T < 5\%$ ). If the upper bound of the 95% central posterior credible interval is below 5%, it will be concluded that there is 95% probability that the investigational lens is statistically significantly lower than 5% based on observed sample.

Bayesian Estimation and Statistical Evaluation of Hypothesis:

The null and alternative hypotheses for unacceptable lens fitting of the investigational lens compared to the threshold of 20% are as follows:

$$H_o: p_T \ge 20\%$$
  
 $H_1: p_T < 20\%$ 

where  $p_T$  is the probability of an unacceptable lens fitting across all study visits for test lens. Based on Bayesian posterior probability distribution of the proportion  $p_T$ , superiority is interpreted as 95% probability of test being statistically lower than the threshold of 20% (i.e.,  $p_T < 20\%$ ). If the upper bound of the 95% central posterior credible interval is below 20%, it will be concluded that there is 95% probability that the investigational lens is statistically significantly lower than 20% based on observed sample.

In the case of zero clinically significant SLF (or unacceptable lens fitting), a Bayesian hierarchical model accounting for zero-event problem will be considered <sup>16</sup>.

### 14.6. Secondary Analyses

### CLUE Vision, Comfort and, Handling

Secondary endpoints for CLUE vision, comfort and handling, scores after 2-weeks of lens wear will be analyzed separately using the same model as described above for primary analysis of CLUE vision scores.

The null and alternative hypothesis to test for superiority of the hyperopic subjects relative to the pre-defined threshold of 46 for the investigational lens is as follows:

$$H_o$$
:  $\mu_{Hyperopes} \le 46$   
 $H_A$ :  $\mu_{Hyperopes} > 46$ 

Where  $\mu_{Hyperopes}$  represents the population mean for the investigational lens after 2-weeks lens wear with respect to CLUE handling scores for hyperopic subjects. The Test lens will be declared statistically significantly greater than 46 if the one-sided p-values is below 0.025.

The null and alternative hypothesis to test for superiority of the hyperopic subjects relative to the pre-defined threshold of 38 for the investigational lens is as follows:

$$H_o$$
:  $\mu_{Hyperopes} \le 38$   
 $H_A$ :  $\mu_{Hyperopes} > 38$ 

Where  $\mu_{Hyperopes}$  represents the population mean for the investigational lens after 2-weeks lens wear with respect to CLUE comfort scores for hyperopic subjects. The Test lens will be declared statistically significantly greater than 38 if the one-sided p-values is below 0.025.

The null and alternative hypothesis to test for superiority of the myopic subjects relative to the pre-defined threshold of 55 for the investigational lens is as follows:

$$H_o$$
:  $\mu_{Myopes} \le 55$   
 $H_A$ :  $\mu_{Myopes} > 55$ 

Where  $\mu_{Myopes}$  represents the population mean for the investigational lens after 2-weeks lens wear with respect to CLUE handling scores for myopic subjects. The investigational lens will be declared statistically significantly greater than 55 if the one-sided p-values is below 0.025.

The null and alternative hypothesis to test for superiority of the hyperopic subjects relative to the pre-defined threshold of 41 for the Test lens is as follows:

$$H_o$$
:  $\mu_{Hyperopes} \le 41$   
 $H_A$ :  $\mu_{Hyperopes} > 41$ 

Where  $\mu_{Hyperopes}$  represents the population mean for the investigational lens after 2-weeks lens wear with respect to CLUE vision scores for hyperopic subjects. The investigational lens will be declared statistically significantly greater than 41 if the one-sided p-values is below 0.025.

The null and alternative hypothesis to test for superiority of the myopic subjects relative to the pre-defined threshold of 51 for the investigational lens is as follows:

$$H_o$$
:  $\mu_{Myopes} \le 51$   
 $H_A$ :  $\mu_{Myopes} > 51$ 

Where  $\mu_{Myopes}$  represents the population mean for the investigational lens after 2-weeks lens wear with respect to CLUE comfort scores for myopic subjects. The investigational lens will be declared statistically significantly greater than 51 if the one-sided p-values is below 0.025.

The null and alternative hypothesis to test for superiority of the myopic subjects relative to the pre-defined threshold of 46 for the investigational lens is as follows:

$$H_o$$
:  $\mu_{Myopes} \le 46$   
 $H_A$ :  $\mu_{Myopes} > 46$ 

Where  $\mu_{Myopes}$  represents the population mean for the investigational lens after 2-weeks lens wear with respect to CLUE vision scores for myopic subjects. The Test lens will be declared statistically significantly greater than 46 if the one-sided p-values is below 0.025.

# Lens Fit Success (Number of lenses required to achieve lens optimization)

Number of lenses required to achieve lens optimization will be analyzed using a Bayesian beta-binomial model with correlated binary data<sup>14</sup>.

### Bayesian Estimation and Statistical Evaluation of Hypothesis:

Superiority of the Test lens relative to the pre-defined threshold with respect to unacceptable lens fitting will be evaluated using Bayesian statistics. The null and alternative hypotheses for evaluating superiority of the investigational lens relative to 90% are as follows:

$$H_0: p_T \le 90\%$$
  
 $H_A: p_T > 90\%$ ,

where  $p_{\rm T}$  is the probability of event (i.e., proportion of subjects to achieve optimization in 4 lenses or less while wearing the test lens). Based on Bayesian posterior probability distribution of the proportion  $p_T$ , superiority is interpreted as 95% probability of the Test lens being statistically greater than the pre-defined threshold of 90% (i.e.,  $p_T > 0.90$ ) with respect to unacceptable lens fitting rate. If the upper bound of the 95% central posterior credible interval is above 0.90, it can be concluded that there is 95% probability that the investigational lens is superior to the 90% threshold (statistically better) based on the observed sample.

In the event that all subjects' vision was optimized in 4 lenses (2 pairs) or less (i.e., zero optimization events), a Bayesian hierarchical model accounting for zero event problem will be considered<sup>16</sup>.

# 14.7. Exploratory Analyses

Not Applicable.

### 14.8. Interim Analysis

Not Applicable.

# 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing values will not be imputed. The count of missing values will be included in the summary tables and listings. Subjects who drop-out early may be replaced to ensure that at least 140 subjects complete the study.

### 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

#### 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

### 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using an EDC system (Clario). An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJVC database manager and sent to JJVC for analysis.

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Only specifically delegated staff can enter data on a CRF. Once completed, the eCRFs will be reviewed for accuracy and completeness and signed by the Investigator. The sponsor or sponsor's representatives will be authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and

confidentiality. After the final database lock, the Investigator will be provided with Individual Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2011.

### 15.2. Subject Record

At a minimum, subject record should be available for the following:

- subject identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication
- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is considered to be the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

### 15.3. Trial Registration on ClinicalTrials.gov

This study will be registered on ClinicalTrials.gov based on the following: The purpose of the study is for design confirmation, not feasibility.

### 16. DATA MANAGEMENT

#### 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJVC must be contacted and notified in writing within 24 hours.

### 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJVC. The Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJVC will use information developed in this clinical study in connection with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she has an obligation to provide complete test results and all data developed during this study to the Sponsor.

### 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, include the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJVC may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source data/documents and reports for the purpose of monitoring and auditing by JJVC and for inspection by local and regulatory authorities.

#### 16.4. Data Monitoring Committee

Not applicable.

### 17. CLINICAL MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent versions, and regulatory requirements are maintained.
- Ensuring the rights and wellbeing of subjects are protected.
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel.
- Ensuring that protocol deviations are documented with corrective action plans, as applicable.

- Ensuring that the clinical site has sufficient test article and supplies.
- Clarifying questions regarding the study.
- Resolving study issues or problems that may arise.
- Reviewing of study records and source documentation verification in accordance with the monitoring plan.

#### 18. ETHICAL AND REGULATORY ASPECTS

### 18.1. Study-Specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study, and during the study, subjects will be given any new information that may affect their decision to continue participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Only subjects who are fully able to understand the risks, benefits, and potential adverse events of the study, and provide their consent voluntarily will be enrolled.

### 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, ISO14155:2020<sup>1</sup>, and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64<sup>th</sup> WMA General Assembly 2013<sup>2</sup> and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with applicable regulatory requirements.

#### 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol.
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information).
- Sponsor-approved subject recruitment materials.
- Information on compensation for study-related injuries or payment to subjects for participation in the study.
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB).
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects.
- Any other documents that the IEC/IRB requests to fulfill its obligation.

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, the informed consent form, applicable recruiting materials, and subject compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study, the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol revisions
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- If applicable, new or revised subject recruitment materials approved by the Sponsor
- Revisions to compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's Brochure revisions
- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)
- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol revisions that increase subject risk, the revisions and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

### 18.4. Informed Consent

Each subject or their representative, must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki<sup>2</sup>, ISO14155:2020<sup>1</sup> guidelines, applicable regulatory requirements, and Sponsor Policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

The subject will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the subject.

### 18.5. Privacy of Personal Data

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Health Information Portability and Accountability Act (HIPAA) in the United States<sup>17</sup> and other applicable personal data protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and subject records.

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations.

The Sponsor ensures that the personal data will be:

- processed fairly and lawfully.
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes.
- adequate, relevant, and not excessive in relation to said purposes.
- accurate and, where necessary, kept current.

Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential.

#### 19. STUDY RECORD RETENTION

In compliance with the ISO 14155:2020<sup>1</sup> guidelines, the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ISO 14155:2020<sup>1</sup> and all study documents as specified by the applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least two (2) years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least two (2) years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports. If the Investigator has a question regarding retention of study records, he/she should contact JJVC.

#### 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Clinical Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJVC management representative prior to study initiation.

JJVC reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible subject in the study.
- Scheduling a study visit outside the subject's acceptable visit range.

JJVC reserves the right to withhold final remuneration until all study related activities have been completed, such as:

- Query resolution.
- Case Report Form signature.
- Completion of any follow-up action items.

#### 21. PUBLICATION

There is no plan to publish the outcome of this investigation, but the study sponsor may choose to publish study results if this is needed to support future regulatory submissions or marketing activities.

#### 22. REFERENCES

- 1 ISO 14155:2020: Clinical investigation of medical devices for human subjects Good clinical practice, Available at: https://www.iso.org/standard/71690.html
- 2 Declaration of Helsinki Ethical principles for Medical Research Involving Human Subjects, Available at: https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/
- 3 United States (US) Code of Federal Regulations (CFR). Available at: https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR
- 4 Franklin R. Investigator's Brochure CR-6542, v1.0 ( ): Evaluation of the clinical performance of Daily Disposable Silicone Hydrogel Multifocal Toric Contact Lenses.
- 6 Franklin R. Clinical Study Protocol , v6. ( ). Evaluation of Silicone Hydrogel Multifocal Toric Contact Lenses in a Hyperopic Population. January 11, 2021.
- 7 Franklin R. Clinical Study Protocol , v1. ( ). Evaluation of Daily Disposable Silicone Hydrogel Multifocal Toric Contact Lenses. May 12, 2021.
- 8 Franklin R. Clinical Study Protocol , v1.0 ( ). Evaluation of Rotation with a Multifocal Toric Contact Lens. June 02, 2022.

- 9 Wirth RJ, Edwards MC, Henderson M, Henderson T, Olivares G, Houts CR. Development of the contact lens user experience: CLUE scales . *Optometry and Vision Science*. 2016;93(8):801. Available at: https://pubmed.ncbi.nlm.nih.gov/27383257/
- 10 Project Aurora for Astigmatism Customer Requirements Document (CRD),
- 11 SAS Institute Inc: SAS® 9.4 Statements: Reference, Third Edition. Cary, NC SAS Institute Inc; 2014.
- 12 Cannon J. Technical Report Post-Marketing CLUE Scores Analysis of Toric and Multifocal Toric CL Wearers. April 14, 2022.
- 13 PASS. Power Analysis and Sample Size Software. Kaysville, Utah, USA: NCSS, LLC; 2021. https://www.ncss.com/software/pass/pass-documentation
- 14 Diniz CAR, Tutia MH, Leite JG. Bayesian analysis of a correlated binomial model. *Brazilian Journal of Probability and Statistics*. 2010;24(1):68-77.
- 15 Kenward MG, Roger JH. Small Sample Inference for Fixed Effects from Restricted Maximum Likelihood. *Biometrics*. 1997;53(3):983-997.
- 16 Jovanovic BD. and Levy PS. A Look at the Rule of Three. *The American Statistician*. 1997;51(2):137-139.
- 17 Health Information Portability and Accountability Act (HIPAA), Available at: https://www.hhs.gov/hipaa/for-professionals/privacy/index.html

APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES)



Page 87 of 171































# **APPENDIX B: PATIENT INSTRUCTION GUIDE**

Will be provided separately.

# APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT)

Not Applicable, as this study uses Investigational Products
APPENDIX D: LENS FITTING GUIDE







#### APPENDIX E: PRESBYOPIC SYMPTOMS QUESTIONNAIRE



#### APPENDIX F: OCULAR DOMINANCE



#### APPENDIX G: BINOCULAR OVER REFRACTION



#### APPENDIX H:

- DETERMINATION OF NEAR ADDITION
  NEAR logMAR VISUAL ACUITY MEASUREMENT PROCEDURE
  LENS FITTING CHARACTERISTICS
  SUBJECT REPORTED OCULAR SYMPTOMS
  DETERMINATION OF DISTANCE SPHEROCYLINDRICAL
  - REFRACTIONS
- BIOMICROSCOPY SCALE
- KERATOMETRY
- DISTANCE AND NEAR VISUAL ACUITY EVALUATION
- TORIC FIT EVALUATION
- ETDRS DISTANCE VISUAL ACUITY MEASURMENT PROCEDURE
- VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION

**TESTING** 



**Document Type:** 

Document Number: Revision Number: 5

NEAR LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE





| Title: | <b>Lens Fitting Char</b> | racteristics |
|------------------------|--------------------------|--------------------|
| <b>Document Type:</b> | | |
| <b>Document Number</b> | • | Revision Number: 6 |

Document Type:

Document Number: 6







DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS



BIOMICROSCOPY SCALE






**Biomicroscopy Scale** Title: **Document Type: Document Number:** Revision Number: 10


Title: **Biomicroscopy Scale Document Type: Document Number:** Revision Number: 10







| Title: | Keratometry Procedure | | |
|---|---|---|---|
| Document Type:<br>Document Number: | | Revision Number: | 03 |
| _ | | | |

DISTANCE AND NEAR VISUAL ACUITY EVALUATION

**Document Type:** 

Document Number: 5







Document Type:
Document Number: **Revision Number: 7** 



DISTANCE LOGMAR VISUAL ACUITY MESAUREMENT PROCEDURE



Page 2 of 3



VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION TESTING

Document Number: Revision Number: 4

Title: Visual Acuity Chart Luminance and Room Illumination Testing **Document Type: Document Number: Revision Number: 4**  Title:

| Γitle: | Visual Acuity C | Acuity Chart Luminance and Room Illumination Testing |
|---|---|---|
| Document Type: | | |
| Document Number: | | Revision Number: 4 |



#### PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

Protocol Number and Title: CR-6542 Evaluation of the clinical performance of Daily Disposable Silicone Hydrogel Multifocal Toric Contact Lenses

Version and Date: 4.0, 25 March 2024

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to ISO 14155:2020<sup>1</sup>, the Declaration of Helsinki<sup>2</sup>, United States (US) Code of Federal Regulations (CFR)<sup>3</sup>, and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. I, as the Principal Investigator, am responsible for ensuring that all clinical site personnel, including Sub-Investigators, adhere to all regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

| Principal Investigator: | | |
|-------------------------|------------------------------------------|------|
| | Signature | Date |
| | Name and Professional Position (Printed) | - |
| Institution/Site: | | |
| | Institution/Site Name | |
| | Institution/Site Address | |